CLINICAL TRIAL: NCT02928224
Title: A Multicenter, Randomized, Open-label, 3-Arm Phase 3 Study of Encorafenib + Cetuximab Plus or Minus Binimetinib vs. Irinotecan/Cetuximab or Infusional 5-Fluorouracil (5-FU)/Folinic Acid (FA)/Irinotecan (FOLFIRI)/Cetuximab With a Safety Lead-in of Encorafenib + Binimetinib + Cetuximab in Patients With BRAF V600E-mutant Metastatic Colorectal Cancer
Brief Title: Study of Encorafenib + Cetuximab Plus or Minus Binimetinib vs. Irinotecan/Cetuximab or Infusional 5-Fluorouracil (5-FU)/Folinic Acid (FA)/Irinotecan (FOLFIRI)/Cetuximab With a Safety Lead-in of Encorafenib + Binimetinib + Cetuximab in Patients With BRAF V600E-mutant Metastatic Colorectal Cancer
Acronym: BEACON CRC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry); Pierre Fabre Medicament (Industry); Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-818-302; BEACON CRC (Other: Alias Study Number); 2015-005805-35 (EudraCT Number); C4221009 (Other: Pfizer)
Record Dates: First submitted 2016-08-16; First posted 2016-10-10 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: BRAF V600E-mutant Metastatic Colorectal Cancer
Keywords: Colorectal cancer; BRAF; BRAFV600E
MeSH Terms: conditions — Colorectal Neoplasms | interventions — encorafenib; binimetinib; Cetuximab; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (3):
- Safety Lead-in, Triplet Arm (Experimental): Encorafenib + binimetinib + cetuximab.
  Interventions: Drug: Encorafenib; Drug: Binimetinib; Drug: Cetuximab
- Doublet Arm (Experimental): Encorafenib + cetuximab.
  Interventions: Drug: Encorafenib; Drug: Cetuximab
- Control Arm (Active Comparator): Investigator's choice of either irinotecan/cetuximab or FOLFIRI/cetuximab.
  Interventions: Drug: Cetuximab; Drug: Irinotecan; Drug: Folinic Acid; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Encorafenib — Orally, once daily.
  Arms: Doublet Arm; Safety Lead-in, Triplet Arm
Drug: Binimetinib — Orally, twice daily.
  Arms: Safety Lead-in, Triplet Arm
Drug: Cetuximab — Standard of care.
Drug: Irinotecan — Standard of care.
  Arms: Control Arm
Drug: Folinic Acid — Standard of care.
  Other Names: FA
  Arms: Control Arm
Drug: 5-Fluorouracil — Standard of care.
  Other Names: 5-FU
  Arms: Control Arm

SUMMARY:
This is a multicenter, randomized, open-label, 3-arm Phase 3 study to evaluate encorafenib + cetuximab plus or minus binimetinib versus Investigator's choice of either irinotecan/cetuximab or FOLFIRI/cetuximab, as controls, in patients with BRAFV600E mCRC whose disease has progressed after 1 or 2 prior regimens in the metastatic setting. The study contains a Safety Lead-in Phase in which the safety and tolerability of encorafenib + binimetinib + cetuximab will be assessed prior to the Phase 3 portion of the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years at time of informed consent
* Histologically- or cytologically-confirmed CRC that is metastatic
* Presence of BRAFV600E in tumor tissue as previously determined by a local assay at any time prior to Screening or by the central laboratory
* Progression of disease after 1 or 2 prior regimens in the metastatic setting
* Evidence of measurable or evaluable non-measurable disease per RECIST, v1.1
* Adequate bone marrow, cardiac, kidney and liver function
* Able to take oral medications
* Female patients are either postmenopausal for at least 1 year, are surgically sterile for at least 6 weeks, or must agree to take appropriate precautions to avoid pregnancy from screening through follow-up if of childbearing potential
* Males must agree to take appropriate precautions to avoid fathering a child from screening through follow-up

Key Exclusion Criteria:

* Prior treatment with any RAF inhibitor, MEK inhibitor, cetuximab, panitumumab or other epidermal growth factor receptor (EGFR) inhibitors
* Prior irinotecan hypersensitivity or toxicity that would suggest an inability to tolerate irinotecan 180 mg/m2 every 2 weeks
* Symptomatic brain metastasis or leptomeningeal disease
* History or current evidence of retinal vein occlusion or current risk factors for retinal vein occlusion (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes)
* Known history of acute or chronic pancreatitis
* History of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) ≤12 months prior to randomization
* Uncontrolled blood pressure despite medical treatment
* Impaired GI function or disease that may significantly alter the absorption of encorafenib or binimetinib (e.g., ulcerative diseases, uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption)
* Concurrent or previous other malignancy within 5 years of study entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in-situ of the cervix, or other noninvasive or indolent malignancy
* History of thromboembolic or cerebrovascular events ≤ 6 months prior to starting study treatment, including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis or pulmonary emboli
* Concurrent neuromuscular disorder that is associated with the potential of elevated creatine (phosphor)kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* Residual common terminology criteria for adverse events (CTCAE) ≥ Grade 2 toxicity from any prior anticancer therapy, with the exception of Grade 2 alopecia or Grade 2 neuropathy
* Known history of HIV infection
* Active hepatitis B or hepatitis C infection
* Known history of Gilbert's syndrome
* Known contraindication to receive cetuximab or irinotecan at the planned doses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2019-02-11 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (411):
- United States (89):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - Compassionate Care Research Group, Inc. at Compassionate Cancer Care Medical Group, Inc., Fountain Valley, California
  - Keck Hospital of USC - Norris Healthcare Center (HC3), Los Angeles, California
  - Keck Hospital of USC, Los Angeles, California
  - LAC+USC Medical Center, Los Angeles, California
  - Norris Healthcare Center 3 (HC3), Los Angeles, California
  - USC Eye Institute, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Harvard Eye Associates, Orange, California
  - Rocky Mountain Lions Eye Institute, Aurora, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado Denver CTO (CTRC), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - University of Colorado Hospital Inpatient Pavillion', Aurora, Colorado
  - Smilow Cancer Hospital at Yale - New Haven, New Haven, Connecticut
  - Temple Medical Center, New Haven, Connecticut
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center at North Haven, North Haven, Connecticut
  - The Lennar Foundation Medical Center, Coral Gables, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Dr. Clayton Berger (opthalmology), Fort Lauderdale, Florida
  - Mehmet F. Hepgur, MD - Broward Health Medical Center, Fort Lauderdale, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center/UMHC, Miami, Florida
  - Sylvester at Kendall, Miami, Florida
  - Illinois CancerCare- Bloomington, Bloomington, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Illinois CancerCare- Galesburg, Galesburg, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - The University of Chicago Medicine Center for Advanced Care Orland Park, Orland Park, Illinois
  - Illinois CancerCare- Ottawa, Ottawa, Illinois
  - Illinois Cancer Care, PC, Peoria, Illinois
  - Illinois Eye Center, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Investigational Drug Services IUHSCC, Indianapolis, Indiana
  - Sidney &Lois Eskenazi Hospital, Indianapolis, Indiana
  - IU Health Springmill, Indianapolis, Indiana
  - Baptist Health Floyd Cancer Center, New Albany, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - The University of Kansas Hospital, Kansas City, Kansas
  - KU Eye, Prairie Village, Kansas
  - The University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - The University of Kansas Cancer Center, Investigational Drug Services, Westwood, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - The Investigational Drug Pharmacy (IDS) in the Sidney Kimmel Cancer Center at Johns Hopkins, Baltimore, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Ophthalmic Consultants of Boston Inc, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Siteman Cancer Center - St Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Saint Louis University, St Louis, Missouri
  - Washington University Infusion Center Pharmacy, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Memorial Sloan Kettering: Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering: Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering: Rockefeller Outpatient Pavilion, New York, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - Casey Eye Institute-South Waterfront, Portland, Oregon
  - OHSU Center for Health and Healing, Portland, Oregon
  - OHSU Research Pharmacy Services, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Scott & White Clinic - Temple Pavilion, Temple, Texas
  - Scott & White Medical Center - Temple, Temple, Texas
  - Spokane Eye Clinic, Spokane, Washington
  - Inland Imaging, LLC Holy Family Hospital, Spokane, Washington
  - Medical Oncology Associates, PS DBA Summit Cancer Centers, Spokane, Washington
  - Providence Holy Family Nuclear Medicine, Spokane, Washington
  - Medical Oncology Associates, PS DBA Summit Cancer Centers, Spokane Valley, Washington
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
- Argentina (5):
  - CLINICA PERGAMINO S.A. (Centro de Investigacion Pergamino S.A.), Pergamino, Buenos Aires
  - Centro Medico INFINITO, Santa Rosa, La Pampa Province
  - Centro Medico CAIPO (Centro para la Atención del paciente Oncológico), San Miguel de Tucumán, Tucumán Province
  - Clinica Universitaria Reina Fabiola, Córdoba
  - Centro Oncologico Riojano Integral - CORI, La Rioja
- Australia (11):
  - St Vincent's Clinic, Darlinghurst, NEW South Wales (nsw)
  - St Vincent's Hospital Sydney, Darlinghurst, NEW South Wales (nsw)
  - Marsden Eye Specialists, Parramatta, NEW South Wales (nsw)
  - Newcastle Eye Centre, Sydney, NEW South Wales (nsw)
  - Mater Misericordiae Limited, South Brisbane, Queensland
  - Central Adelaide Local Health Network Inc. operating as Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Central Adelaide Local Health Network Inc. operating as The Queen Elizabeth Hospital, Woodville South, South Australia
  - Monash Health Translation Precinct - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Austria (9):
  - Klinikum Wels - Grieskirchen GmbH, Abteilung fuer Innere Medizin IV, Wels, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH, Abteilung fuer Augenheilkunde und Optometrie, Wels, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH, Abteilung fuer Innere Medizin II, Wels, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH, Institut fuer Nuklearmedizin, Wels, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH, Institut fuer Radiologie I, Wels, Upper Austria
  - DZU, Diagnose Zentrum Urania GmbH, Vienna
  - AKH Wien, Vienna
  - Medizinische Universitaet Wien/AKH Wien, Vienna
  - Medizinische Universität Wien/AKH Wien, Vienna
- Belgium (11):
  - Centre Hospitalier de l'Ardenne - Site de Libramont, Libramont-Chevigny, Luxembourg
  - AZ Sint-Jan Brugge - Oostende AV - Campus Sint-Jan - Oncology, Bruges, WEST Vlaanderen
  - Imelda Ziekenhuis, Bonheiden
  - Grand Hopital de Charleroi (GHdC), Charleroi
  - UZ Antwerpen, Edegem
  - AZ Maria Middelares, Ghent
  - University Hospital Gasthuisberg (UZ Leuven), Leuven
  - Centre Hospitalier Universitaire (CHU) de Liege, Liège
  - CHC Saint Joseph, Liège
  - AZ Delta Roeselaere-Menen, Roeselaere
  - Centre Hospitalier Regional (CHR) - Verviers, Verviers
- Brazil (39):
  - CEMES Centro Medico Especializado em Oftalmologia, Cachoeiro de Itapemirim, Espírito Santo
  - Centro de Pesquisas Clínicas em Oncologia, Cachoeiro de Itapemirim, Espírito Santo
  - Hospital Evangelico de Cachoeiro de Itapemirim, Cachoeiro de Itapemirim, Espírito Santo
  - Hospital do Olho, Salvador, Estado de Bahia
  - CENOB - Centro de Oncologia da Bahia SS Ltda / Oncovida, Salvador, Estado de Bahia
  - Instituto Vizibelli, Belo Horizonte, Minas Gerais
  - CENANTRON - Centro Avancado de Tratamento Oncologic, Belo Horizonte, Minas Gerais
  - Fundação Universidade de Caxias do Sul, Caxias do Sul, Rio Grande do Sul
  - Daniel Lubisco Pandolfi, Lajeado, Rio Grande do Sul
  - Sociedade Beneficencia e Cardade de Lajeado/Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Associacao Hospitalar Beneficente Sao Vicente de Paulo / Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Consultorio Medico de Oftalmologia - Dr. Ricardo Tres, Passo Fundo, Rio Grande do Sul
  - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Thiago Vernetti Ferreira, Pelotas, Rio Grande do Sul
  - Leandro Becker, Pelotas, Rio Grande do Sul
  - Fernanda Mendes, Pelotas, Rio Grande do Sul
  - UPCO - Unidade de Pesquisas Clinicas em Oncologia, Pelotas, Rio Grande do Sul
  - Fernanda Lauermann, Pelotas, Rio Grande do Sul
  - Diogo Duarte Torre, Porto Alegre, Rio Grande do Sul
  - Farmacia Central da Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Nucleo de Novos Tratamentos em Cancer, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clínica de Oncologia e Hematologia - Hospital Mãe de Deus/AESC, Porto Alegre, Rio Grande do Sul
  - Clinica de Oftalmologia Lavinsky, Porto Alegre, Rio Grande do Sul
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Giuliano Santos Borges - ME / Clinica de Neoplasias Litoral - Centro de Novos Tratamentos Itajai, Itajaí, Santa Catarina
  - Clinica Toller, Barretos, São Paulo
  - Olhos Centro Diagnostico e Laser LTDA, Barretos, São Paulo
  - Fundacao Pio XII, Barretos, São Paulo
  - FUNDAÇÃO DO ABC - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - CEPOS - Centro de Estudos e Pesquisas Oncologicas de Sorocaba, Sorocaba, São Paulo
  - Instituto de Oncologia de Sorocaba "Dr. Gilson Delgado", Sorocaba, São Paulo
  - Karen Miyuki Kubokawa Shorer, Sorocaba, São Paulo
  - Oftalmologia Diagnostica de Sorocaba (ODS), Sorocaba, São Paulo
  - Instituto de Ensino e Pesquisa São Lucas, São Paulo
  - Instituto de Ensino e Pesquisa São Lucas - Pharmacy, São Paulo
  - Hospital Leforte, São Paulo
  - IPEPO - Instituto da Visao, São Paulo
- Canada (6):
  - Eye Care Centre, Vancouver General Hospital, Vancouver, British Columbia
  - BC Cancer, Vancouver Center, Vancouver, British Columbia
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Centre integre universitaire de sante et de services sociaux de l'Ouest-de-l'Ile-de-Montreal, Montreal, Quebec
- Chile (2):
  - Instituto Clinico Oncologico del Sur (ICOS), Temuco, Región de la Araucanía
  - Hospital Clinico Vina Del Mar, Viña del Mar, V Region Valparaiso
- Czechia (12):
  - Ocni ordinace Oftalpro s.r.o., Brno
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fingerlanduv ustav patologie, Hradec Králové
  - I. interni kardioangiologicka klinika, Hradec Králové
  - Klinika nemoci koznich a pohlavnich, Hradec Králové
  - Nemocnicni lekarna - Usek klinickych studii, Hradec Králové
  - Ocni klinika, Hradec Králové
  - Radiologicka klinika, Hradec Králové
  - Fakultni nemocnice Olomouc, I. interni klinika - kardiologicka, Olomouc
  - Fakultni nemocnice Olomouc, Lekarna, Olomouc
  - Fakultni nemocnice Olomouc, Olomouc
- Odense University Hospital (OUH), Odense C, Denmark
- France (15):
  - Hopital Jean Minjoz, Besançon
  - CHU Morvan, Brest
  - Centre Ophtalmologique - Pole Vision - Clinique Val d'Ouest, Écully
  - Centre Leon Berard, Lyon
  - ICM Val d'Aurelle, Montpellier
  - CHU HOTEL-Dieu, Nantes
  - Hopital Georges Pompidou, Paris
  - Centre hospitalier national d'ophtalmologie des Quinze-Vingts, Paris
  - Centre Hospitalier National d'Opthalmologie des Quinze-Vingts (CHNO des XV-XX), Paris
  - CHU Robert Debre, Reims
  - SCM Centre d'ophtalmologie, Saint Jeand de Vedas
  - CHU Toulouse - Purpan, hopital Pierre-Paul Riquet, Toulouse
  - CHU Toulouse-Institut Inuversitaire du Cancer Toulouse, Toulouse
  - CHU Toulouse-Rangueil, Toulouse
  - Gustave Roussy, Villejuif
- Germany (33):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Augenklinik der Universitaet Muenchen, Munich, Bavaria
  - LMU Klinikum der Universitaet Muenchen, Campus Grosshadern, Munich, Bavaria
  - Augenarzt-Gemeinschaftspraxis Dr.med.Andreas Kind & Dr.med. Ute Kariger-Schweigert, Falkensee, Brandenburg
  - Medizinische Hochschule Hannover (MHH), Hanover, Lower Saxony
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Institut f. Pathologie - Ruhr-Universitaet Bochum, Prof. Dr. med. Andrea Tannapfel, Bochum, North Rhine Westfalia
  - Kliniken Essen Mitte / Knappschaftskrankenhaus, Essen, North Rhine-Westphalia
  - Praxis fuer Augenheilkunde Dr. Edmund Meyer-Schwickerath, Essen, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Essen, North Rhine-Westphalia
  - Universitaetsklinikum Essen (AoeR), Innere Klinik (Tumorforschung), Westdeutsches Tumorzentrum, Essen, North Rhine-Westphalia
  - Universitaetsklinikum Essen; Diagnostischeu. Interventionelle Radiologie u. Neuroradiologie, Essen, North Rhine-Westphalia
  - Universitaetsklinikum Essen; Nuklearmedizin, Essen, North Rhine-Westphalia
  - Universitaetsklinikum Essen; Zentralapotheke, Essen, North Rhine-Westphalia
  - Evang. Krankenhaus Essen - Werden; Klinik fuer Augenheilkunde, Essen, North Rhine-Westphalia
  - Augentagesklinik Maria-Hilf Krankenhaus, Mönchengladbach, North Rhine-Westphalia
  - Kliniken Maria Hilf GmbH - Franziskuskrankenhaus, Mönchengladbach, North Rhine-Westphalia
  - Kliniken Maria Hilf GmbH; Klinik fuer Radiologie, Mönchengladbach, North Rhine-Westphalia
  - Lukaskrankenhaus Neuss; Zentrale Apotheke, Neuss, North Rhine-Westphalia
  - Augenarzt Praxis Dr. med. Petra Huelsmann, Worms, Rhineland-Palatinate
  - Gemeinschaftspraxis fuer Radiologie und Nuklearmedizin, Standort Worms, Worms, Rhineland-Palatinate
  - Martin Apotheke, Worms, Rhineland-Palatinate
  - Onkologische Schwerpunktpraxis Worms, Worms, Rhineland-Palatinate
  - Praxisgemeinschaft Kruse + Hofstaetter, Worms, Rhineland-Palatinate
  - Evangelisches Waldkrankenhaus Spandau, Berlin
  - Universitaetsklinikum Carl Gustav Carus der Technischen Universitaet Dresden, Dresden
  - Universitaetsklinikum Hamburg Eppendorf, Klinik fuer Augenheilkunde, Hamburg
  - Facharztzentrum Eppendorf, Hamburg
  - Universitaetsklinikum Hamburg Eppendorf, Zentrum fuer Radiologie und Endoskopie, Hamburg
  - ZytoService Deutschland GmbH, Standort-Hamburg-Jenfeld, Hamburg
  - HKS Kardiologische Praxis am Israelitischen Krankenhaus, Hamburg
  - Radiologie im Israelitischen Krankenhaus, Hamburg
- Hungary (9):
  - Zala Megyei Szent Rafael Korhaz - Onkologiai Osztaly, Zalaegerszeg, Zala County
  - Szent Margit Kórház, Budapest
  - Eszak-Pesti Centrumkorhaz-Honvedkorhaz, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Egyesitett Szent Istvan es Szent Laszlo Korhaz-Rendelointezet, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Pecsi Tudomanyegyetem Altalanos Orvostudomanyi Kar, Pécs
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
- Israel (13):
  - Tel Aviv Sourasky Medical Center - Oncology, Tel Aviv, NAP
  - The Barzilai Medical Center - Oncology Institute, Ashkelon
  - Soroka University Medical Center, Beersheba
  - MOR Institute, Bnei Brak
  - Ein-Karem Department of Medical Imaging of Hadassah Medical Organization, Hadassah Medical Center,, Jerusalem
  - Hadassah Medical Organization, Hadassah Medical Center, Ein-Karem, Jerusalem
  - Pharmacy of Hadassah Medical Organization, Hadassah Medical Center, Ein-Karem, Jerusalem
  - Mt. Scopus Department of Medical Imaging of Hadassah Medical Organization,, Jerusalem
  - Imaging Department of Meir Medical Center, Kfar Saba
  - Meir Medical Center, Kfar Saba
  - Pharmacy of Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (40):
  - Ospedali Riuniti Umberto I, Torrette Di Ancona, Ancona
  - ASST Bergamo Ovest, Ospedale Treviglio Caravaggio di Trevigl, Treviglio, Bergamo
  - Oculistica, ASST Papa Giovanni XXIII, Bergamo, BG
  - Oncologia, ASST Papa Giovanni XXIII, Bergamo, BG
  - Clinica di Oncologia Medica AOU di Cagliari Presidio Duilio Casula Monserrato, Monserrato, Cagliari
  - Farmacia AOU di Cagliari Presidio Duilio Casula Monserrato, Monserrato, Cagliari
  - Radiologia AOU di Cagliari Presidio Duilio Casula Monserrato, Monserrato, Cagliari
  - Oculistica - ASST Cremona, Ospedale di Cremona, Cremona, CR
  - SC Farmacia Aziendale - ASST Cremona, Ospedale di Cremona, Cremona, CR
  - SC Oncologia - ASST Cremona, Ospedale di Cremona, Cremona, CR
  - U.O. Oculistica, Istituto Clinico HUMANITAS, Rozzano, Milano
  - U.O. di Oncologia ed Ematologia, Istituto Clinico HUMANITAS, Rozzano (MI), Milan
  - IRCCS Ospedale San Raffaele - U.O. di Medicina Oncologica, Milan, MI
  - Servizio di Farmacia - IRCCS Ospedale San Raffaele, Milan, MI
  - S.C. Radiologia diagnostica e interventistica - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - SC Oncologia Medica 1, SS Oncologia Medica Gastroenterologica, Milan, MI
  - Cardiologia per i pazienti oncologici - Istituto Oncologico Veneto I.R.C.C.S, Padua, PD
  - Clinica Oculistica - Azienda Ospedaliera di Padova, Padua, PD
  - U.O. Oncologia Medica 1 - Istituto Oncologico Veneto I.R.C.C.S, Padua, PD
  - Policlinico S.Orsola Malpighi, AOU di Bologna - Oncologia Medica, Bologna
  - Divisione Anatomia Patologica Presidio San Giovanni di Dio, Cagliari
  - Oculistica AOU di Cagliari Presidio San Giovanni di Dio, Cagliari
  - Dipartimento Neuromuscoloscheletrico e Organi di Senso, "Oncologia Oculare Unit", Florence
  - SC oncologia Medica I - Azienda Ospedaliero Universitaria Careggi, Florence
  - Radiologia, Milan
  - Unita di Oncologia Medica Gastrointestinale e Tumori Neuroendocrini, Milan
  - Grande Ospedale Metropolitano Niguarda, Milan
  - Dipartimento Interaziendale Farmaceutico - AOU Policlinico di Modena, Modena
  - SC di Oftalmologia - AOU Policlinico di Modena, Modena
  - SC di Radiologia, Dipartimento Interaziendale integrato Diagnostica per Immagini, Modena
  - SSD Day Hospital Oncologico - Dipartimento ad attivita integrata di Oncologia, Ematologia, Modena
  - AOU Universita degli Studi della Campania L. Vanvitelli - DAI di Medicina Interna e Specialistica, Napoli
  - AOU Universita degli Studi della Campania L. Vanvitelli - U. Ma.Ca., Napoli
  - AOU Universita degli Studi della Campania L. Vanvitelli, Napoli
  - UO Oculistica - AOU Pisana, Stabilimento Ospedaliero di Cisanello, Pisa
  - SOD Radiodiagnostica 3 - AOU Pisana, Stabilimento Ospedaliero di Santa Chiara, Pisa
  - UO Farmaceutica, Gestione del Farmaco - AOU Pisana, Stabilimento Ospedaliero di Santa Chiara, Pisa
  - UO Oncologia Medica 2 - AOU Pisana, Stabilimento Ospedaliero di Santa Chiara, Pisa
  - U.O.S.D. Oncologia Medica, Dipartimento di Medicina - Fondazione PTV Policlinico Tor Vergata, Roma
  - U.O.S.D. Patologie Retiniche - Fondazione PTV Policlinico Tor Vergata, Roma
- Japan (13):
  - Chayagasaka Eye Clinic, Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Tsukahara Eye Clinic, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Osaka University Hospital Laboratory for Clinical Investigation, Suita, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyushu Central Hospital of the Mutual Aid Association of Public School Teachers, Fukuoka
  - National Hospital Organization Osaka National Hospital, Osaka
- Mexico (2):
  - Consultorio dentro de la Torre Medica Dalinde (Oncologia Medica), Mexico City, Cuauhtemoc
  - Superare Centro de Infusion S.A. de C.V., Delegacion Cuauhtemoc, Mexico City
- Netherlands (7):
  - Rijnstate Hospital Arnhem, Arnhem, Gelderland
  - Rijnstate Hospital Velp, Velp, Gelderland
  - Maastricht University Medical Center (MUMC), Maastricht, Limburg
  - The Netherlands Cancer Institute, Amsterdam, North Holland
  - Onze Lieve Vrouwen Gasthuis, Amsterdam, North Holland
  - Haga Ziekenhuis, The Hague, South Holland
  - Universitair Medisch Centrum Utrecht, Utrecht
- Norway (4):
  - Colosseum Øyelegesenter C/O LB Holdings AS, Lommedalen
  - Colosseum Øyelegesenter C/O LB Holdings AS, Oslo
  - Oslo universitetssykehus, Radiumhospitalet, Oslo
  - Sykehusapoteket Oslo, Radiumhospitalet, Oslo
- Poland (7):
  - Szpital Specjalistyczny W Brzozowie, Podkarpacki Osrodek Onkologiczny Im.Ks.B.Markiewicza, Brzozów
  - Wojewodzki Szpital Zespolony, Oddzial Onkologiczny, Elblag
  - Szpital Specjalistyczny im. L. Rydygiera w Krakowie Sp.z.o.o., Krakow
  - Europejskie Centrum Zdrowia Otwock, Szpital im. F. Chopina, Otwock
  - NZOZ Centrum Medyczne HCP, Poznan
  - NZOZ Przychodnia Specjalistyczna GUTMED, Poznan
  - MAGODENT Sp. z o.o. Szpital Elblaska, Warsaw
- Russia (6):
  - Regional Budgetary Healthcare Institution Kursk Regional Clinical, Kursk, Kursk Oblast
  - Evimed Llc, Chelyabinsk
  - Federal State Budget Institution "N.N. Blokhin Russian Cancer Research Center" of the, Moscow
  - Federal State Budget Institution "N.N. Blokhin Russian Cancer Research Center", Moscow
  - A. Tsyb Medical Radiological Research Center - branch of the, Obninsk
  - State Budgetary Educational Institution of Higher Professional Education First Saint Petersburg, Saint Petersburg
- South Korea (13):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Anyang, Gyeonggido
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Korea University Guro Hospital, Seoul, Seoul Teugbyeolsi
  - Dong-A University Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital IRB, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (30):
  - Complejo Hospitalario de Jaen, Jaén, Andalusia
  - Sercosa - Clinica de las Nieves, Jaén, Andalusia
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Institut Catala d'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba, Cordona
  - Hospital Nuestra Señora del Rosario, Madrid, Madrid, Communidad Delaware
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital del Mar, Barcelona
  - Clinica Corachan, Barcelona
  - Hospital Quiron Salud Barcelona, Barcelona
  - Cetir Centre Medic S.L., Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Consulta Dr. Juan Carlos Castillo Dominguez, Córdoba
  - Gabinete Radiologico Dr. Pita, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital HM Universitario Sanchinarro, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Clinica Oftalvist, Valencia
  - Fundacion Instituto Valenciano de Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Quiron Salud Zaragoza, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (6):
  - Changhua Christian Hospital, Changhua, Changhua County
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- Turkey (Türkiye) (7):
  - Ege University Medical Faculty, Izmir, Bornova
  - Izmir Medical Park Hospital - Medical Oncology, Izmir, Izmir, Karsiyaka
  - Medeniyet University Goztepe Training and Research Hospital, Istanbul, Kadikoy
  - Hacettepe University Medical Faculty, Ankara
  - Uludag University Hospital, Bursa
  - Trakya Universitesi Tip Fakultesi, Edirne
  - Inonu Universitesi Turgut Ozal Medical Center, Malatya
- Ukraine (12):
  - Oftalmolohycheskyi tsentr "Vzghliad" MTs, Dnipropetrovsk, Dnipropetrovsk Oblast
  - Derzhavnyi zaklad, Dnipropetrovska medychna akademiia Ministerstva okhorony zdorovia Ukrainy, Dnipropetrovsk, Dnipropetrovsk Oblast
  - Komumalnyi zaklad, Dnipropetrovska miska bahatoprofilna klinichna likarnia Nº4, Dnipropetrovsk, Dnipropetrovsk Oblast
  - Kyivska klinichna likarnia na zaliznychnomu transporti No3 filii Tsentr okhorony zdorov'ia PAT, Kyiv, Kyivska Oblast'
  - Natsionalnyi medychnyi universytet imeni O.O Bohomltsia, kafedra onkolohii, Kyiv, Kyivska Oblast'
  - Natsionalnyi medychnyi universytet imeni O.O Bohomltsia, kafedra oftalmolohii, Kyiv, Kyivska Oblast
  - Oleksandrivska klinichna likarnia mista Kyieva, Kyiv, Kyivska Oblast
  - Kyivskyi miskyi klinichnyi onkotsentr, Kyiv, Kyivska Oblast
  - Vinnytskyi oblasnyi klinichnyi onkolohichnyi dyspanser, viddilennia khimioterapii, Vinnytsia, Vinnytsia Oblast
  - DVNZ "Uzhhorodskyi natsionalnyi universytet", Uzhhorod, Zakarpattia Oblast
  - TOV "Zakarpatskyi Tsentr Mikrokhirurhii Oka", Uzhhorod, Zakarpattia Oblast
  - Tsentralna miska klinichna likarnia, Miskyi onkolohichnyi tsentr, Uzhhorod, Zakarpattia Oblast
- United Kingdom (9):
  - NHS Grampian - Aberdeen Royal Infirmary, Aberdeen, Aberdeenshire Scotland
  - King Edward V11 Hospital, Windsor, Berkshire
  - Beatson West of Scotland Cancer Centre, Glasglow, Glasglow City, Scotland
  - University Hospitals Birmingham NHS Foundation Trust Queen Elizabeth Hospital, Birmingham, WEST Midlands
  - Hammersmith Hospital, Imperial College Healthcare NHS Trust, London
  - Imperial College Healthcare NHS Trust, Hammersmith Hospital, London
  - Sarah Cannon Research Institute UK, London
  - Imperial College Healthcare NHS Trust, Charing Cross Hospital, London
  - The Christie NHS Foundation Trust - Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Kopetz S, Murphy DA, Pu J, Ciardiello F, Desai J, Van Cutsem E, Wasan HS, Yoshino T, Saffari H, Zhang X, Hamilton P, Xie T, Yaeger R, Tabernero J. Molecular profiling of BRAF-V600E-mutant metastatic colorectal cancer in the phase 3 BEACON CRC trial. Nat Med. 2024 Nov;30(11):3261-3271. doi: 10.1038/s41591-024-03235-9. Epub 2024 Sep 23. PMID 39313594
- [Derived] Taieb J, Lonardi S, Desai J, Folprecht G, Gallois C, Marques EP, Khan S, Castagne C, Wasan H. Adverse Events Associated with Encorafenib Plus Cetuximab in Patients with BRAFV600E-mutant Metastatic Colorectal Cancer: An in-depth Analysis of the BEACON CRC Study. Clin Colorectal Cancer. 2023 Mar;22(1):59-66. doi: 10.1016/j.clcc.2022.12.003. Epub 2022 Dec 24. PMID 36653241
- [Derived] Stintzing S, Seufferlein T, Rose C, Reichenbach F, Luftner D. Encorafenib in Combination With Cetuximab After Systemic Therapy in Patients With BRAFV600E Mutant Metastatic Colorectal Cancer: German Health Technology Assessment-Driven Analyses From the BEACON CRC Study. Clin Colorectal Cancer. 2022 Sep;21(3):244-251. doi: 10.1016/j.clcc.2022.04.002. Epub 2022 May 5. PMID 35654691
- [Derived] Kopetz S, Grothey A, Van Cutsem E, Yaeger R, Wasan H, Yoshino T, Desai J, Ciardiello F, Loupakis F, Hong YS, Steeghs N, Guren TK, Arkenau HT, Garcia-Alfonso P, Belani A, Zhang X, Tabernero J. Quality of life with encorafenib plus cetuximab with or without binimetinib treatment in patients with BRAF V600E-mutant metastatic colorectal cancer: patient-reported outcomes from BEACON CRC. ESMO Open. 2022 Jun;7(3):100477. doi: 10.1016/j.esmoop.2022.100477. Epub 2022 May 30. PMID 35653981
- [Derived] Tabernero J, Grothey A, Van Cutsem E, Yaeger R, Wasan H, Yoshino T, Desai J, Ciardiello F, Loupakis F, Hong YS, Steeghs N, Guren TK, Arkenau HT, Garcia-Alfonso P, Elez E, Gollerkeri A, Maharry K, Christy-Bittel J, Kopetz S. Encorafenib Plus Cetuximab as a New Standard of Care for Previously Treated BRAF V600E-Mutant Metastatic Colorectal Cancer: Updated Survival Results and Subgroup Analyses from the BEACON Study. J Clin Oncol. 2021 Feb 1;39(4):273-284. doi: 10.1200/JCO.20.02088. PMID 33503393
- [Derived] Kopetz S, Grothey A, Yaeger R, Van Cutsem E, Desai J, Yoshino T, Wasan H, Ciardiello F, Loupakis F, Hong YS, Steeghs N, Guren TK, Arkenau HT, Garcia-Alfonso P, Pfeiffer P, Orlov S, Lonardi S, Elez E, Kim TW, Schellens JHM, Guo C, Krishnan A, Dekervel J, Morris V, Calvo Ferrandiz A, Tarpgaard LS, Braun M, Gollerkeri A, Keir C, Maharry K, Pickard M, Christy-Bittel J, Anderson L, Sandor V, Tabernero J. Encorafenib, Binimetinib, and Cetuximab in BRAF V600E-Mutated Colorectal Cancer. N Engl J Med. 2019 Oct 24;381(17):1632-1643. doi: 10.1056/NEJMoa1908075. Epub 2019 Sep 30. PMID 31566309
- [Derived] Van Cutsem E, Huijberts S, Grothey A, Yaeger R, Cuyle PJ, Elez E, Fakih M, Montagut C, Peeters M, Yoshino T, Wasan H, Desai J, Ciardiello F, Gollerkeri A, Christy-Bittel J, Maharry K, Sandor V, Schellens JHM, Kopetz S, Tabernero J. Binimetinib, Encorafenib, and Cetuximab Triplet Therapy for Patients With BRAF V600E-Mutant Metastatic Colorectal Cancer: Safety Lead-In Results From the Phase III BEACON Colorectal Cancer Study. J Clin Oncol. 2019 Jun 10;37(17):1460-1469. doi: 10.1200/JCO.18.02459. Epub 2019 Mar 20. PMID 30892987
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=ARRAY-818-302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were at least 18 years of age with confirmed metastatic colorectal cancer (CRC) whose disease had progressed after 1 or 2 prior regimens in the metastatic setting and whose tumor tissue was BRAF V600E-mutant as previously determined by a local assay at any time prior to Screening.
Groups:
- Combined Safety Lead-in; Phase 3: Triplet Arm: Encorafenib + binimetinib + cetuximab. Encorafenib: Orally, once daily. Binimetinib: Orally, twice daily. Cetuximab: Standard of care.
- Phase 3: Doublet Arm: Encorafenib + cetuximab. Encorafenib: Orally, once daily. Cetuximab: Standard of care.
- Phase 3: Control Arm: Investigator's choice of either irinotecan/cetuximab or FOLFIRI/cetuximab. Cetuximab: Standard of care. Irinotecan: Standard of care. Folinic Acid: Standard of care. 5-Fluorouracil: Standard of care. Following protocol amendment, eligible participants could crossover to receive either triplet or doublet regimen.
Period: Overall Study
Arm/Group | Combined Safety Lead-in | Phase 3: Triplet Arm | Phase 3: Doublet Arm | Phase 3: Control Arm
Started | 37 | 224 | 220 | 221
Crossover Participants | 0 | 0 | 0 | 3 (Participants from control arm received triplet therapy.)
Completed | 0 | 0 | 0 | 0
Not Completed | 37 | 224 | 220 | 221
Not completed — Lost to Follow-up | 1 | 1 | 3 | 0
Not completed — Death | 30 | 209 | 193 | 198
Not completed — Withdrawal by Subject | 0 | 3 | 7 | 20
Not completed — Study participation terminated by sponsor | 3 | 8 | 12 | 3
Not completed — Other | 3 | 3 | 5 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consists of the Full Analysis Set (FAS). For participants in the CSLI, the FAS includes all participants who received at least 1 dose of study drug and had at least 1 post treatment assessment, which may include death. For the randomized Phase 3 portion of the study, the FAS consists of all randomized participants.
Groups:
- Combined Safety Lead-in (CSLI); Phase 3: Triplet Arm: Encorafenib + binimetinib + cetuximab. Encorafenib: Orally, once daily. Binimetinib: Orally, twice daily. Cetuximab: Standard of care.
- Total: Total of all reporting groups
Arm/Group | Combined Safety Lead-in (CSLI) | Phase 3: Triplet Arm | Phase 3: Doublet Arm | Phase 3: Control Arm | Total
Number analyzed (Participants) | 37 | 224 | 220 | 221 | 702
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 141 | 137 | 149 | 450
  >=65 years | 14 | 83 | 83 | 72 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (10.34) | 59.5 (11.65) | 60.2 (11.65) | 58.4 (12.07) | 59.3 (11.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 119 | 106 | 127 | 374
  Male | 15 | 105 | 114 | 94 | 328
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 14 | 13 | 6 | 33
  Not Hispanic or Latino | 37 | 203 | 195 | 202 | 637
  Unknown or Not Reported | 0 | 7 | 12 | 13 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 7 | 20 | 25 | 39 | 91
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 0 | 3
  White | 29 | 195 | 183 | 172 | 579
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 7 | 11 | 10 | 28
Region [Count of Participants; unit: Participants]
  North America | 5 | 30 | 28 | 29 | 92
  Europe | 25 | 150 | 145 | 125 | 445
  Rest of World | 7 | 44 | 47 | 67 | 165
Eastern Cooperative Oncology Group Performance Status (ECOG PS) at Baseline [Count of Participants; unit: Participants] — ECOG PS was used to assess the physical health of participants, and ranges from 0 to 5 where 0: fully active, 1: restricted in physically strenuous activity, 2: ambulatory and capable of self-care but unable to work, 3: capable only of limited self-care , 4: completely disabled; cannot carry on any self-care; totally confined to bed or chair, 5: dead.
  Participants
    0-Fully active | 22 | 116 | 112 | 108 | 358
    1-Restircted in physically strenuous activity | 15 | 108 | 104 | 113 | 340
    2-Ambulatory and capable of all self-care | 0 | 0 | 4 | 0 | 4
Number of Participants According to Primary Tumor Location [Count of Participants; unit: Participants]
  Left Colon | 11 | 79 | 83 | 68 | 241
  Right Colon | 23 | 126 | 110 | 119 | 378
  Left and Right Colon | 0 | 8 | 11 | 22 | 41
  Unknown | 3 | 11 | 16 | 12 | 42
Number of Participants According to Removal of Primary Tumor [Count of Participants; unit: Participants]
  Completely Resected | 20 | 133 | 123 | 122 | 398
  Partially Resected/Unresected | 17 | 91 | 97 | 99 | 304
Number of Participants According to Number of Organs Involved [Count of Participants; unit: Participants]
  <=2 | 16 | 114 | 117 | 123 | 370
  3+ | 21 | 110 | 103 | 98 | 332
Sites of Metastases [Number; unit: Sites] — One participant may have more than one site of metastases.
  Sites
    Liver | 24 | 145 | 134 | 128 | 431
    Lung | 10 | 86 | 83 | 86 | 265
    Lymph Node | 17 | 86 | 82 | 88 | 273
    Peritoneum/Omentum | 17 | 77 | 97 | 93 | 284

OUTCOME MEASURES:

1. Primary Outcome: (Safety Lead-in) Number of Participants With Dose-Limiting Toxicities (DLTs)
Time Frame: Cycle 1 (up to 28 days)
Population: The dose-determining set (DDS) consisted of all CSLI participants from the safety set who either completed a minimum exposure requirement (received >= 75% dose intensity of the planned dose for each binimetinib, encorafenib and cetuximab) and had sufficient safety evaluations or experienced a dose-limiting toxicity (DLT).
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Safety Lead-in (CSLI)
Number analyzed (Participants) | 37
Participants | 5

2. Primary Outcome: (Safety Lead-in) Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. Number of participants reporting AEs were reported in this outcome measure.
Time Frame: Duration of safety lead-in, approximately 6 months (up to 28 days per cycle)
Population: The safety set consisted of all participants who received at least 1 dose of study drug and had at least 1 post-treatment assessment, which may have included death. Participants were analyzed according to treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Participants | 37

3. Primary Outcome: (Safety Lead-in) Incidence of Dose Interruptions, Dose Modifications and Discontinuations Due to Adverse Events (AEs) - Interim Analysis
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. Number of participants with dose interruptions, dose modifications and dose discontinuations due to AEs were reported in this outcome measure.
Time Frame: Duration of safety lead-in, approximately 6 months (up to 28 days per cycle)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Participants | 26

4. Primary Outcome: (Safety Lead-in) Incidence of Dose Interruptions, Dose Modifications and Discontinuations Due to Adverse Events (AEs) - Final Analysis
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. Number of participants according to incidence of dose interruptions, dose modifications and dose discontinuations due to AEs were reported in this outcome measure.
Time Frame: From start of study treatment until 30 days post last dose of study treatment (maximum treatment exposure of 280 weeks)
Population: The safety set consisted of all participants who received at least 1 dose of study drug and had at least 1 posttreatment assessment, which may have included death. Participants were analyzed according to treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Participants
  Dose interruptions | 30
  Dose modifications | 16
  Discontinuation due to AEs | 8

5. Primary Outcome: (Phase 3) Overall Survival (OS) of Triplet Arm vs. Control Arm - Interim Analysis
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: From randomization to death due to any cause until 204 deaths were observed (maximum treatment exposure of 89.1 weeks for triplet arm and 52.4 weeks for control arm)
Population: The Full Analysis Set (FAS) for the Phase 3 portion of the study consisted of all randomized Phase 3 participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Triplet Arm | Phase 3: Control Arm
Number analyzed (Participants) | 224 | 221
Months | 9.03 [8.02 to 11.43] | 5.42 [4.76 to 6.57]
Statistical Analysis 1: Comparison: Phase 3: Triplet Arm vs Phase 3: Control Arm; Test type: Other; p < 0.0001, Stratified Log-rank

6. Other Pre Specified Outcome: (Phase 3) Overall Survival (OS) of Triplet Arm vs. Control Arm - Final Analysis
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: From randomization to death due to any cause (maximum treatment exposure of 277.4 weeks for triplet arm and 108 weeks for control arm)
Population: The FAS for the Phase 3 portion of the study consisted of all randomized Phase 3 participants.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase 3:Control Arm: Investigator's choice of either irinotecan/cetuximab or FOLFIRI/cetuximab. Cetuximab: Standard of care. Irinotecan: Standard of care. Folinic Acid: Standard of care. 5-Fluorouracil: Standard of care. Following protocol amendment, eligible participants could crossover to receive either triplet or doublet regimen.
Arm/Group | Phase 3: Triplet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 224 | 221
Months | 9.82 [8.34 to 11.73] | 5.88 [5.09 to 7.16]
Statistical Analysis 1: Comparison: Phase 3: Triplet Arm vs Phase 3:Control Arm; Test type: Other; p < 0.0001, Stratified Log-rank

7. Primary Outcome: (Phase 3) Objective Response Rate (ORR) by Blinded Independent Central Review (BICR) Per Response Evaluation Criteria in Solid Tumors (RECIST), v1.1 of Triplet Arm vs. Control Arm
Description: ORR per RECIST, v1.1, was defined as the percentage of participants achieving an overall best response of complete response (CR) or partial response (PR), where CR: disappearance of all target and non-target lesions and normalization of tumor marker level, all lymph nodes must be non-pathological in size (<10 millimeter [mm] short axis), and PR: at least 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters persistence of one or more non-target lesions and/or maintenance of tumor marker level above the normal limits.
Time Frame: Duration of Phase 3, approximately 6 months (up to 28 days per cycle)
Population: The Phase 3 Response Efficacy Set consisted of the first 330 participants randomized into the Phase 3 portion of the study and any additional participants randomized on the same day as the 330th randomized participant.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 3: Triplet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 111 | 107
Percentage of participants | 26.1 [18.2 to 35.3] | 1.9 [0.2 to 6.6]
Statistical Analysis 1: Comparison: Phase 3: Triplet Arm vs Phase 3:Control Arm; Test type: Other; p < 0.0001, Chi-squared

8. Secondary Outcome: (Safety Lead-in) Objective Response Rate (ORR) by Investigator
Description: ORR per RECIST, v1.1, was defined as the percentage of participants achieving an overall best response of CR or PR, where CR: disappearance of all target and non-target lesions and normalization of tumor marker level, all lymph nodes must be non-pathological in size (<10 mm short axis), and PR: at least 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters persistence of one or more non-target lesions and/or maintenance of tumor marker level above the normal limits.
Time Frame: From start of study treatment until 30 days post last dose of study treatment (maximum treatment exposure of 280 weeks)
Population: The Safety Lead-in (SLI) Efficacy Set consisted of all CSLI participants in the FAS who were identified at screening as having a BRAF V600E mutation (per local or central testing).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 36
Percentage of participants | 52.8 [35.5 to 69.6]

9. Secondary Outcome: (Safety Lead-in) Objective Response Rate (ORR) by BICR
Description: as for outcome 8
Time Frame: From start of study treatment until 30 days post last dose of study treatment (maximum treatment exposure of 280 weeks)
Population: The SLI Efficacy Set consisted of all CSLI participants in the FAS who were identified at screening as having a BRAF V600E mutation (per local or central testing).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 36
Percentage of participants | 41.7 [25.5 to 59.2]

10. Secondary Outcome: (Safety Lead-in) Duration of Response (DOR) by Investigator
Description: DOR was defined as the time from first radiographic evidence of response to the earliest documented disease progression (PD) or death due to underlying disease. PD: at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions were evaluated.
Time Frame: From time of response to the earliest documented PD or death due to underlying disease (maximum treatment exposure of 280 weeks)
Population: The SLI Efficacy Set consisted of all CSLI participants in the FAS who were identified at screening as having a BRAF V600E mutation (per local or central testing). Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 19
Months | 6.47 [4.17 to 11.07]

11. Secondary Outcome: (Safety Lead-in) Duration of Response (DOR) by BICR
Description: DOR was defined as the time from first radiographic evidence of response to the earliest documented PD or death due to underlying disease. PD: at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions were evaluated.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 15
Months | 8.15 [2.79 to NA] — NA= not reached. Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval.

12. Secondary Outcome: (Safety Lead-in) Time to Response by Investigator
Description: Time to response was defined as the time from first dose to first radiographic evidence of response.
Time Frame: From first dose to first radiographic evidence of response (maximum treatment exposure of 280 weeks)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 36
Months | 1.45 [1.38 to 1.64]

13. Secondary Outcome: (Safety Lead-in) Time to Response by BICR
Description: Time to response was defined as the time from first dose to first radiographic evidence of response.
Time Frame: From first dose to first radiographic evidence of response (maximum treatment exposure of 280 weeks)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 36
Months | 1.45 [1.38 to 1.64]

14. Secondary Outcome: (Safety Lead-in) Progression-Free Survival (PFS) by Investigator
Description: PFS was defined as the time from first dose to the earliest documented PD or death due to any cause. PD: at least a 20% increase (including an absolute increase of at least 5 mm) in the sum of diameters of target lesions, taking as reference the smallest sum on study and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions were evaluated.
Time Frame: From first dose to the earliest documented PD or death due to any cause (maximum treatment exposure of 280 weeks)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 36
Months | 8.08 [5.59 to 9.3]

15. Secondary Outcome: (Safety Lead-in) Progression-Free Survival (PFS) by BICR
Description: as for outcome 14
Time Frame: From first dose to the earliest documented PD or death due to any cause (maximum treatment exposure of 280 weeks)
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 36
Months | 5.59 [4.44 to 9.3]

16. Secondary Outcome: (Phase 3) Overall Survival (OS) in Doublet Arm vs. Control Arm
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: From randomization to death due to any cause until 204 deaths were observed (maximum treatment exposure of 89.7 weeks for doublet arm and 52.4 weeks for control arm)
Population: The FAS for the Phase 3 portion of the study consisted of all randomized Phase 3 participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Doublet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 220 | 221
Months | 9.40 [8.11 to 11.24] | 5.88 [5.09 to 7.16]
Statistical Analysis 1: Comparison: Phase 3: Doublet Arm vs Phase 3:Control Arm; Test type: Other; p < 0.0001, Stratified Log-rank

17. Secondary Outcome: (Phase 3) Overall Survival (OS) in Triplet Arm vs. Doublet Arm
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: From randomization to death due to any cause until 204 deaths were observed (maximum treatment exposure of 89.7 weeks for doublet arm and 89.1 weeks for triplet arm)
Population: The FAS for the Phase 3 portion of the study consisted of all randomized Phase 3 participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Triplet Arm | Phase 3: Doublet Arm
Number analyzed (Participants) | 224 | 220
Months | 9.82 [8.34 to 11.73] | 9.40 [8.11 to 11.24]
Statistical Analysis 1: Comparison: Phase 3: Triplet Arm vs Phase 3: Doublet Arm; Test type: Other; p = 0.5958, Stratified Log-rank

18. Secondary Outcome: (Phase 3) Comparison of Progression-Free Survival (PFS) in Triplet Arm vs Control Arm Per BICR
Description: as for outcome 14
Time Frame: From first dose to the earliest documented PD or death due to any cause (maximum treatment exposure of 277.4 weeks for triplet arm and 108 weeks for control arm)
Population: The FAS for the Phase 3 portion of the study consisted of all randomized Phase 3 participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Triplet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 224 | 221
Months | 4.30 [4.14 to 5.19] | 1.51 [1.45 to 1.71]
Statistical Analysis 1: Comparison: Phase 3: Triplet Arm vs Phase 3:Control Arm; Test type: Other; p < 0.0001, Stratified Log-rank

19. Secondary Outcome: (Phase 3) Comparison of Progression-free Survival (PFS) in Triplet Arm vs Control Arm Per Investigator
Description: as for outcome 14
Time Frame: as for outcome 18
Population: The FAS for the Phase 3 portion of the study consisted of all randomized Phase 3 participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Triplet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 224 | 221
Months | 4.47 [4.24 to 5.36] | 1.58 [1.51 to 2.07]
Statistical Analysis 1: Comparison: Phase 3: Triplet Arm vs Phase 3:Control Arm; Test type: Other; p < 0.0001, Stratified Log-rank

20. Secondary Outcome: (Phase 3) Comparison of Progression-Free Survival (PFS) in Doublet Arm vs Control Arm Per BICR
Description: as for outcome 14
Time Frame: From first dose to the earliest documented PD or death due to any cause (maximum treatment exposure of 268 weeks for doublet arm and 108 weeks for control arm)
Population: The FAS for the Phase 3 portion of the study consisted of all randomized Phase 3 participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Doublet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 220 | 221
Months | 4.21 [3.71 to 5.36] | 1.51 [1.45 to 1.71]
Statistical Analysis 1: Comparison: Phase 3: Doublet Arm vs Phase 3:Control Arm; Test type: Other; p < 0.0001, Stratified Log-rank

21. Secondary Outcome: (Phase 3) Comparison of Progression-Free Survival (PFS) in Doublet Arm vs Control Arm Per Investigator
Description: as for outcome 14
Time Frame: as for outcome 20
Population: The FAS for the Phase 3 portion of the study consisted of all randomized Phase 3 participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Doublet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 220 | 221
Months | 4.27 [4.04 to 5.36] | 1.58 [1.51 to 2.07]
Statistical Analysis 1: Comparison: Phase 3: Doublet Arm vs Phase 3:Control Arm; Test type: Other; p < 0.0001, Stratified Log-rank

22. Secondary Outcome: (Phase 3) Comparison of Progression-Free Survival (PFS) in Triplet Arm vs Doublet Arm Per BICR
Description: as for outcome 14
Time Frame: From first dose to the earliest documented PD or death due to any cause (maximum treatment exposure of 277.4 weeks for triplet arm and 268 weeks for doublet arm)
Population: The FAS for the Phase 3 portion of the study consisted of all randomized Phase 3 participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Triplet Arm | Phase 3: Doublet Arm
Number analyzed (Participants) | 224 | 220
Months | 4.30 [4.14 to 5.19] | 4.21 [3.71 to 5.36]
Statistical Analysis 1: Comparison: Phase 3: Triplet Arm vs Phase 3: Doublet Arm; Test type: Other; p = 0.1004, Stratified Log-rank

23. Secondary Outcome: (Phase 3) Comparison of Progression-Free Survival (PFS) in Triplet Arm vs Doublet Arm Per Investigator
Description: as for outcome 14
Time Frame: as for outcome 22
Population: The FAS for the Phase 3 portion of the study consisted of all randomized Phase 3 participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Triplet Arm | Phase 3: Doublet Arm
Number analyzed (Participants) | 224 | 220
Months | 4.47 [4.24 to 5.36] | 4.27 [4.04 to 5.36]
Statistical Analysis 1: Comparison: Phase 3: Triplet Arm vs Phase 3: Doublet Arm; Test type: Other; p = 0.3724, Stratified Log-rank

24. Secondary Outcome: (Phase 3) Comparison of Objective Response Rate (ORR) in Triplet Arm vs Control Arm Per Investigator
Description: as for outcome 8
Time Frame: Duration of Phase 3, approximately 6 months (up to 28 days per cycle)
Population: The Phase 3 Response Efficacy Set consisted of the first 330 participants randomized into the Phase 3 portion of the study and any additional participants randomized on the same day as the 330th randomized participant. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 3: Triplet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 111 | 107
Percentage of participants | 26.1 [18.2 to 35.3] | 3.7 [1.0 to 9.3]
Statistical Analysis 1: Comparison: Phase 3: Triplet Arm vs Phase 3:Control Arm; Test type: Other; p < 0.0001, Chi-squared

25. Secondary Outcome: (Phase 3) Comparison of Objective Response Rate (ORR) in Doublet Arm vs Control Arm Per BICR
Description: as for outcome 8
Time Frame: Duration of Phase 3, approximately 6 months (up to 28 days per cycle)
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 3: Doublet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 113 | 107
Percentage of participants | 20.4 [13.4 to 29.0] | 1.9 [0.2 to 6.6]
Statistical Analysis 1: Comparison: Phase 3: Doublet Arm vs Phase 3:Control Arm; Test type: Other; p < 0.0001, Chi-squared

26. Secondary Outcome: (Phase 3) Comparison of Objective Response Rate (ORR) in Doublet Arm vs Control Arm Per Investigator
Description: as for outcome 8
Time Frame: Duration of Phase 3, approximately 6 months (up to 28 days per cycle)
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 3: Doublet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 113 | 107
Percentage of participants | 15.9 [9.7 to 24.0] | 3.7 [1.0 to 9.3]
Statistical Analysis 1: Comparison: Phase 3: Doublet Arm vs Phase 3:Control Arm; Test type: Other; p < 0.0001, Chi-squared

27. Secondary Outcome: (Phase 3) Comparison of Objective Response Rate (ORR) in Triplet Arm vs Doublet Arm Per BICR
Description: as for outcome 8
Time Frame: Duration of Phase 3, approximately 6 months (up to 28 days per cycle)
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 3: Triplet Arm | Phase 3: Doublet Arm
Number analyzed (Participants) | 111 | 113
Percentage of participants | 26.1 [18.2 to 35.3] | 20.4 [13.4 to 29.0]
Statistical Analysis 1: Comparison: Phase 3: Triplet Arm vs Phase 3: Doublet Arm; Test type: Other; p = 0.1928, Cochran-Mantel-Haenszel

28. Secondary Outcome: (Phase 3) Comparison of Objective Response Rate (ORR) in Triplet Arm vs Doublet Arm Per Investigator
Description: as for outcome 8
Time Frame: Duration of Phase 3, approximately 6 months (up to 28 days per cycle)
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 3: Triplet Arm | Phase 3: Doublet Arm
Number analyzed (Participants) | 111 | 113
Percentage of participants | 26.1 [18.2 to 35.3] | 15.9 [9.7 to 24.0]
Statistical Analysis 1: Comparison: Phase 3: Triplet Arm vs Phase 3: Doublet Arm; Test type: Other; p = 0.0357, Cochran-Mantel-Haenszel

29. Secondary Outcome: (Phase 3) Comparison of Duration of Response (DOR) in Triplet Arm vs Control Arm Per BICR
Description: as for outcome 11
Time Frame: From time of response to PD or death due to underlying disease (maximum treatment exposure of 277.4 weeks for triplet arm and 108 weeks for control arm)
Population: as for outcome 24
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Triplet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 111 | 107
Months | 4.80 [2.96 to 9.69] | NA [2.56 to NA] — NA= not reached. Insufficient number of participants with events to calculate the median and upper limit of the 95% confidence interval.

30. Secondary Outcome: (Phase 3) Comparison of Duration of Response (DOR) in Triplet Arm vs Control Arm Per Investigator
Description: as for outcome 10
Time Frame: as for outcome 29
Population: as for outcome 24
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Triplet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 111 | 107
Months | 4.80 [3.29 to 6.57] | 5.75 [2.56 to NA] — NA= not reached. Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval.

31. Secondary Outcome: (Phase 3) Comparison of Duration of Response (DOR) in Doublet Arm vs Control Arm Per BICR
Description: as for outcome 11
Time Frame: From time of response to PD or death due to underlying disease (maximum treatment exposure of 268 weeks for doublet arm and 108 weeks for control arm)
Population: as for outcome 24
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Doublet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 113 | 107
Months | 6.06 [4.07 to 8.28] | NA [2.56 to NA] — NA= not reached. Insufficient number of participants with events to calculate the median and upper limit of the 95% confidence interval.

32. Secondary Outcome: (Phase 3) Comparison of Duration of Response (DOR) in Doublet Arm vs Control Arm Per Investigator
Description: as for outcome 11
Time Frame: as for outcome 31
Population: as for outcome 24
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Doublet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 113 | 107
Months | 5.70 [3.65 to 6.74] | 5.75 [2.56 to NA] — NA= not reached. Insufficient number of participants with events to calculate the upper limit of the 95% confidence interval.

33. Secondary Outcome: (Phase 3) Comparison of Duration of Response (DOR) in Triplet Arm vs Doublet Arm by BICR
Description: as for outcome 11
Time Frame: From time of response to PD or death due to underlying disease (maximum treatment exposure of 277.4 weeks for triplet arm and 268 weeks for doublet arm)
Population: as for outcome 24
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase 3:Doublet Arm: Encorafenib + cetuximab. Encorafenib: Orally, once daily. Cetuximab: Standard of care.
Arm/Group | Phase 3: Triplet Arm | Phase 3:Doublet Arm
Number analyzed (Participants) | 111 | 113
Months | 4.80 [2.96 to 9.69] | 6.06 [4.07 to 8.28]

34. Secondary Outcome: (Phase 3) Comparison of Duration of Response (DOR) in Triplet Arm vs Doublet Arm by Investigator
Description: as for outcome 11
Time Frame: as for outcome 33
Population: as for outcome 24
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Triplet Arm | Phase 3:Doublet Arm
Number analyzed (Participants) | 111 | 113
Months | 4.80 [3.29 to 6.57] | 5.70 [3.65 to 6.74]

35. Secondary Outcome: (Phase 3) Comparison of Time to Response in Triplet Arm vs Control Arm Per BICR
Description: Time to response was defined as the time from first dose to first radiographic evidence of response.
Time Frame: From first dose to first radiographic evidence of response (maximum treatment exposure of 277.4 weeks for triplet arm and 108 weeks for control arm)
Population: The FAS for the Phase 3 portion of the study consisted of all randomized Phase 3 participants. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Triplet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 50 | 3
Months | 1.43 [1.41 to 1.51] | 1.45 [1.41 to 2.63]

36. Secondary Outcome: (Phase 3) Comparison of Time to Response in Triplet Arm vs Control Arm Per Investigator
Description: Time to response was defined as the time from first dose to first radiographic evidence of response.
Time Frame: as for outcome 35
Population: as for outcome 35
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Triplet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 49 | 7
Months | 1.48 [1.41 to 1.51] | 2.63 [1.45 to 2.79]

37. Secondary Outcome: (Phase 3) Comparison of Time to Response in Doublet Arm vs Control Arm Per BICR
Description: Time to response was defined as the time from first dose to first radiographic evidence of response.
Time Frame: From first dose to first radiographic evidence of response (maximum treatment exposure of 268 weeks for doublet arm and 108 weeks for control arm)
Population: as for outcome 35
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Doublet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 36 | 3
Months | 1.48 [1.41 to 1.58] | 1.45 [1.41 to 2.63]

38. Secondary Outcome: (Phase 3) Comparison of Time to Response in Doublet Arm vs Control Arm Per Investigator
Description: Time to response was defined as the time from first dose to first radiographic evidence of response.
Time Frame: as for outcome 37
Population: as for outcome 35
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Doublet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 31 | 7
Months | 1.48 [1.41 to 1.54] | 2.63 [1.45 to 2.79]

39. Secondary Outcome: (Phase 3) Comparison of Time to Response in Triplet Arm vs Doublet Arm Per BICR
Description: Time to response was defined as the time from first dose to first radiographic evidence of response.
Time Frame: From first dose to first radiographic evidence of response (maximum treatment exposure of 277.4 weeks for triplet arm and 268 weeks for doublet arm)
Population: as for outcome 35
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Triplet Arm | Phase 3:Doublet Arm
Number analyzed (Participants) | 50 | 36
Months | 1.43 [1.41 to 1.51] | 1.48 [1.41 to 1.58]

40. Secondary Outcome: (Phase 3) Comparison of Time to Response in Triplet Arm vs Doublet Arm Per Investigator
Description: Time to response was defined as the time from first dose to first radiographic evidence of response.
Time Frame: as for outcome 39
Population: as for outcome 35
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 3: Triplet Arm | Phase 3:Doublet Arm
Number analyzed (Participants) | 49 | 31
Months | 1.48 [1.41 to 1.51] | 1.48 [1.41 to 1.54]

41. Secondary Outcome: (Phase 3) Change From Baseline in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire for Cancer Participants (QLQ-C30) Triplet Arm vs Control Arm, Doublet Arm vs Control, and Triplet vs Doublet
Description: The EORTC QLQ-C30 questionnaire consisted of 30 questions generating 5 functional scores (physical, role, cognitive, emotional, & social); a global health (GH) status/global quality of life scale score; 3 symptom scale scores (fatigue, pain, & nausea & vomiting); & 6 standalone one-item scores that capture additional symptoms (dyspnea, appetite loss, sleep disturbance, constipation, & diarrhea) & perceived financial burden. All items were graded by severity experienced during previous week & used 4-point-scale (1: not at all, 2: a little, 3: quite a bit, 4: very much). The scores were converted to health-related quality of life (HRQoL) scale ranging from 0-100. Higher scores indicating higher response levels (i.e., higher functioning, higher symptom severity).
Time Frame: Baseline, Cycle(C)1 Day(D)1 , C2 D1, C3 D1, C4 D1, C5 D1, C6 D1, C7 D1, C8 D1, C9 D1, C10 D1, C11 D1, C12 D1, C13 D1, C14 D1, C15 D1, C16 D1, C17 D1, C18 D1, C19 D1, C20 D1, C21 D1, C22 D1, C23 D1, End of Treatment, 30 Day Follow Up(each cycle of 28 days)
Population: The FAS for the Phase 3 portion of the study consisted of all randomized Phase 3 participants. Here, 'Number Analyzed' signifies number of participants evaluable for the specified timepoints. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Phase 3: Triplet Arm | Phase 3:Doublet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 224 | 220 | 221
Units on a scale
  Baseline: number analyzed (Participants) | 209 | 201 | 200
  Baseline | 62.8 (22.18) | 60.7 (21.33) | 62.8 (21.82)
  Change at Cycle 1 Day 1: number analyzed (Participants) | 138 | 133 | 120
  Change at Cycle 1 Day 1 | -2.4 (13.44) | -4.3 (16.27) | -3.4 (15.60)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 181 | 180 | 123
  Change at Cycle 2 Day 1 | -1.6 (19.06) | 3.8 (18.46) | -1.9 (22.45)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 148 | 142 | 51
  Change at Cycle 3 Day 1 | 0.7 (18.86) | 3.5 (19.96) | -0.2 (24.07)
  Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 105 | 37
  Change at Cycle 4 Day 1 | 0.2 (15.63) | 4.2 (22.17) | 1.4 (21.65)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 99 | 81 | 26
  Change at Cycle 5 Day 1 | -1.1 (18.66) | 4.3 (22.09) | -2.2 (22.06)
  Change at Cycle 6 Day 1: number analyzed (Participants) | 68 | 60 | 13
  Change at Cycle 6 Day 1 | -4.0 (16.76) | 5.6 (23.25) | -4.5 (19.43)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 47 | 50 | 10
  Change at Cycle 7 Day 1 | -2.5 (16.01) | 4.3 (21.77) | 1.7 (12.30)
  Change at Cycle 8 Day 1: number analyzed (Participants) | 39 | 40 | 7
  Change at Cycle 8 Day 1 | -2.6 (14.83) | 4.2 (16.98) | 0.0 (27.64)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 33 | 31 | 7
  Change at Cycle 9 Day 1 | -5.8 (17.74) | -5.6 (16.44) | -4.8 (12.60)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 23 | 24 | 4
  Change at Cycle 10 Day 1 | -3.3 (17.90) | -2.8 (16.97) | 2.1 (20.83)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 16 | 19 | 1
  Change at Cycle 11 Day 1 | -5.2 (20.38) | 3.9 (15.31) | 33.3 (NA) — Number analyzed is 1 so standard deviation (SD) is not available.
  Change at Cycle 12 Day 1: number analyzed (Participants) | 14 | 18 | 2
  Change at Cycle 12 Day 1 | 0.0 (22.41) | -4.6 (13.77) | 4.2 (53.03)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 9 | 13 | 1
  Change at Cycle 13 Day 1 | 0.0 (20.41) | -3.2 (14.25) | 0.0 (NA) — Number analyzed is 1 so SD is not available.
  Change at Cycle 14 Day 1: number analyzed (Participants) | 7 | 7 | 0
  Change at Cycle 14 Day 1 | -1.2 (24.26) | -6.0 (15.00) |
  Change at Cycle 15 Day 1: number analyzed (Participants) | 7 | 6 | 0
  Change at Cycle 15 Day 1 | 3.6 (33.63) | 2.8 (8.61) |
  Change at Cycle 16 Day 1: number analyzed (Participants) | 5 | 3 | 0
  Change at Cycle 16 Day 1 | -16.7 (42.08) | -5.6 (9.62) |
  Change at Cycle 17 Day 1: number analyzed (Participants) | 3 | 3 | 0
  Change at Cycle 17 Day 1 | -27.8 (20.97) | -2.8 (12.73) |
  Change at Cycle 18 Day 1: number analyzed (Participants) | 1 | 3 | 0
  Change at Cycle 18 Day 1 | -16.7 (NA) — Number analyzed is 1 so SD is not available. | -8.3 (8.33) |
  Change at Cycle 19 Day 1: number analyzed (Participants) | 1 | 2 | 0
  Change at Cycle 19 Day 1 | 0.0 (NA) — Number analyzed is 1 so SD is not available. | -8.3 (11.79) |
  Change at Cycle 20 Day 1: number analyzed (Participants) | 1 | 1 | 0
  Change at Cycle 20 Day 1 | -25 (NA) — Number analyzed is 1 so SD is not available. | -8 (NA) — Number analyzed is 1 so SD is not available. |
  Change at Cycle 21 Day 1: number analyzed (Participants) | 1 | 1 | 0
  Change at Cycle 21 Day 1 | 0.0 (NA) — Number analyzed is 1 so SD is not available. | -16.7 (NA) — Number analyzed is 1 so SD is not available. |
  Change at Cycle 22 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Change at Cycle 22 Day 1 |  | -16.7 (NA) — Number analyzed is 1 so SD is not available. |
  Change at Cycle 23 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Change at Cycle 23 Day 1 |  | 0.0 (NA) — Number analyzed is 1 so SD is not available. |
  Change at End of Treatment: number analyzed (Participants) | 74 | 72 | 79
  Change at End of Treatment | -14.1 (22.66) | -13.1 (21.61) | -15.5 (27.04)
  Change at 30 Day Follow Up: number analyzed (Participants) | 24 | 16 | 21
  Change at 30 Day Follow Up | -17.4 (22.51) | -10.4 (15.96) | -24.6 (24.08)

42. Secondary Outcome: (Phase 3) Change From Baseline in the Functional Assessment of Cancer Therapy-Colon Cancer (FACT-C) in Triplet Arm vs Control Arm, Doublet Arm vs Control, and Triplet vs Doublet
Description: FACT-C= Functional Assessment of Chronic Illness Therapy (FACIT), which assessed HRQoL of cancer participants & participants with other chronic illnesses. It consists of total 36 items (27 items of general version of FACT-C and disease-specific subscale containing 9 CRC-specific items), summarized to 5 subscales: physical well-being (7 items), functional well-being (7 items), social/family well-being (7 items); all 3 subscales range:0-28, emotional well-being (6 items) range: 0-24, colorectal cancer subscale (9 items) range: 0-36; higher subscale score= better QoL. All single-item measures range: 0= 'Not at all' to 4= 'Very much'. Table summarizes functional well-being subscale, individual questions are linearly scaled & combined to form functional well-being subscale score (range 0-28). High score represents better QoL.
Time Frame: Baseline,Cycle (C)1 Day (D)1, C2 D1, C3 D1, C4 D1, C5 D1, C6 D1, C7 D1, C8 D1, C9 D1, C10 D1, C11 D1, C12 D1, C13 D1, C14 D1, C15 D1, C16 D1, C17 D1, C18 D1, C19 D1, C20 D1, C21 D1, C22 D1, C23 D1, End of Treatment, 30 Day Follow Up(each cycle of 28 days)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Phase 3: Triplet Arm | Phase 3:Doublet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 224 | 220 | 221
Units on a scale
  Baseline: number analyzed (Participants) | 211 | 199 | 200
  Baseline | 16.3 (6.22) | 16.2 (5.9) | 16.8 (6.07)
  Change at Cycle 1 Day 1: number analyzed (Participants) | 142 | 130 | 117
  Change at Cycle 1 Day 1 | -0.2 (3.36) | -0.9 (4.06) | -1.4 (3.32)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 183 | 176 | 123
  Change at Cycle 2 Day 1 | -0.3 (4.28) | -0.6 (5.08) | -0.9 (4.48)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 148 | 137 | 50
  Change at Cycle 3 Day 1 | -0.2 (5.15) | -0.2 (5.23) | -0.7 (5.03)
  Change at Cycle 4 Day 1: number analyzed (Participants) | 119 | 105 | 37
  Change at Cycle 4 Day 1 | 0.4 (4.53) | -0.1 (4.66) | -1.8 (6.48)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 100 | 81 | 26
  Change at Cycle 5 Day 1 | 0.7 (6.4) | -0.2 (4.5) | -1.6 (4.58)
  Change at Cycle 6 Day 1: number analyzed (Participants) | 68 | 58 | 13
  Change at Cycle 6 Day 1 | 0.7 (6.05) | 0.6 (4.56) | -1.9 (5.3)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 47 | 49 | 10
  Change at Cycle 7 Day 1 | 0.5 (5.85) | -0.1 (4.70) | -0.5 (5.41)
  Change at Cycle 8 Day 1: number analyzed (Participants) | 40 | 39 | 8
  Change at Cycle 8 Day 1 | 0.9 (6.35) | 0.2 (4.24) | -2.1 (4.97)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 32 | 30 | 7
  Change at Cycle 9 Day 1 | -1.9 (4.32) | -0.8 (3.74) | -2.6 (2.30)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 22 | 24 | 4
  Change at Cycle 10 Day 1 | -1.7 (4.76) | -1.3 (3.59) | 0.5 (4.36)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 17 | 19 | 2
  Change at Cycle 11 Day 1 | -1.5 (4.47) | -0.5 (4.65) | -4.5 (7.78)
  Change at Cycle 12 Day 1: number analyzed (Participants) | 14 | 18 | 2
  Change at Cycle 12 Day 1 | -1.5 (4.93) | -1.1 (4.61) | -4.5 (9.19)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 9 | 13 | 1
  Change at Cycle 13 Day 1 | -2.0 (6.76) | -3.2 (5.34) | -8.0 (NA) — Number analyzed is 1 so SD is not available.
  Change at Cycle 14 Day 1: number analyzed (Participants) | 7 | 7 | 0
  Change at Cycle 14 Day 1 | -2.4 (5.22) | -4.0 (5.74) |
  Change at Cycle 15 Day 1: number analyzed (Participants) | 7 | 6 | 0
  Change at Cycle 15 Day 1 | -2.3 (6.85) | -1.5 (4.72) |
  Change at Cycle 16 Day 1: number analyzed (Participants) | 5 | 3 | 0
  Change at Cycle 16 Day 1 | -4.2 (4.02) | -0.7 (0.58) |
  Change at Cycle 17 Day 1: number analyzed (Participants) | 3 | 3 | 0
  Change at Cycle 17 Day 1 | -6.7 (5.51) | -0.7 (4.51) |
  Change at Cycle 18 Day 1: number analyzed (Participants) | 1 | 3 | 0
  Change at Cycle 18 Day 1 | -5.0 (NA) — Number analyzed is 1 so SD is not available. | -3.0 (4.36) |
  Change at Cycle 19 Day 1: number analyzed (Participants) | 1 | 2 | 0
  Change at Cycle 19 Day 1 | -7.0 (NA) — Number analyzed is 1 so SD is not available. | -6.0 (0.00) |
  Change at Cycle 20 Day 1: number analyzed (Participants) | 1 | 1 | 0
  Change at Cycle 20 Day 1 | -6.0 (NA) — Number analyzed is 1 so SD is not available. | -5.0 (NA) — Number analyzed is 1 so SD is not available. |
  Change at Cycle 21 Day 1: number analyzed (Participants) | 1 | 1 | 0
  Change at Cycle 21 Day 1 | -9.0 | -5.0 |
  Change at Cycle 22 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Change at Cycle 22 Day 1 |  | -12.0 (NA) — Number analyzed is 1 so SD is not available. |
  Change at Cycle 23 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Change at Cycle 23 Day 1 |  | -9.0 (NA) — Number analyzed is 1 so SD is not available. |
  Change at End of Treatment: number analyzed (Participants) | 74 | 73 | 79
  Change at End of Treatment | -2.4 (4.84) | -2.2 (5.14) | -3.1 (6.06)
  Change at 30 Day Follow Up: number analyzed (Participants) | 24 | 16 | 21
  Change at 30 Day Follow Up | -3.5 (6.44) | -0.8 (5.42) | -4.2 (6.41)

43. Secondary Outcome: (Phase 3) Change From Baseline in the EuroQol-5D-5L Visual Analog Scale (EQ-5D-5L VAS) in Triplet Arm vs Control Arm, Doublet Arm vs Control, and Triplet vs Doublet
Description: The EQ-5D-5L contains 1 item for each of 5 dimensions of health-related QoL (i.e., mobility, self-care, usual activities, pain or discomfort and anxiety or depression). Response options for each item varied from having no problems to moderate problems or extreme problems. The EQ-5D-5L (v4.0) is a standardized measure of health utility that provides a single index value for one's health status. The EQ-5D-5L is frequently used for economic evaluations of health care and has been recognized as a valid and reliable instrument for this purpose. The EQ visual analog scale (VAS) is a score that is directly reported by the participant and ranges from 0 to 100 (higher is better quality health).
Time Frame: as for outcome 42
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Phase 3: Triplet Arm | Phase 3:Doublet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 224 | 220 | 221
Units on a scale
  Baseline: number analyzed (Participants) | 210 | 203 | 199
  Baseline | 69.0 (19.03) | 66.5 (19.51) | 68.3 (19.71)
  Change at Cycle 1 Day 1: number analyzed (Participants) | 141 | 135 | 120
  Change at Cycle 1 Day 1 | 0.8 (10.89) | -0.9 (14.09) | -2.1 (15.02)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 183 | 181 | 124
  Change at Cycle 2 Day 1 | 1.4 (14.74) | 1.9 (14.81) | -2.4 (17.20)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 150 | 141 | 52
  Change at Cycle 3 Day 1 | 3.0 (13.94) | 4.2 (17.32) | -1.4 (17.40)
  Change at Cycle 4 Day 1: number analyzed (Participants) | 118 | 105 | 37
  Change at Cycle 4 Day 1 | 4.0 (13.06) | 5.6 (14.87) | -0.4 (15.14)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 99 | 80 | 26
  Change at Cycle 5 Day 1 | 3.3 (14.66) | 5.1 (15.11) | 2.5 (11.17)
  Change at Cycle 6 Day 1: number analyzed (Participants) | 66 | 58 | 13
  Change at Cycle 6 Day 1 | 1.3 (13.33) | 2.9 (16.84) | -3.6 (13.26)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 46 | 47 | 10
  Change at Cycle 7 Day 1 | 1.4 (13.64) | 3.6 (16.71) | 2.4 (7.44)
  Change at Cycle 8 Day 1: number analyzed (Participants) | 39 | 39 | 8
  Change at Cycle 8 Day 1 | 4.1 (10.77) | 2.0 (16.11) | -2.8 (12.95)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 33 | 30 | 7
  Change at Cycle 9 Day 1 | 0.3 (15.16) | -4.0 (12.99) | -8.1 (8.80)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 23 | 23 | 4
  Change at Cycle 10 Day 1 | 0.2 (13.34) | -8.1 (13.68) | -1.8 (2.36)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 17 | 18 | 2
  Change at Cycle 11 Day 1 | 0.2 (13.87) | -0.1 (10.15) | 4.0 (8.49)
  Change at Cycle 12 Day 1: number analyzed (Participants) | 13 | 17 | 2
  Change at Cycle 12 Day 1 | -4.0 (20.11) | -0.6 (11.67) | 1.5 (12.02)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 9 | 12 | 1
  Change at Cycle 13 Day 1 | -3.0 (17.17) | -4.1 (14.41) | -2.0 (NA) — Number analyzed is 1 so SD is not available.
  Change at Cycle 14 Day 1: number analyzed (Participants) | 7 | 7 | 0
  Change at Cycle 14 Day 1 | -4.0 (18.06) | -0.4 (13.99) |
  Change at Cycle 15 Day 1: number analyzed (Participants) | 7 | 6 | 0
  Change at Cycle 15 Day 1 | -3.4 (14.67) | 4.2 (7.36) |
  Change at Cycle 16 Day 1: number analyzed (Participants) | 5 | 3 | 0
  Change at Cycle 16 Day 1 | -10.4 (24.87) | 3.3 (2.89) |
  Change at Cycle 17 Day 1: number analyzed (Participants) | 3 | 3 | 0
  Change at Cycle 17 Day 1 | -18.3 (20.21) | 1.7 (5.77) |
  Change at Cycle 18 Day 1: number analyzed (Participants) | 1 | 3 | 0
  Change at Cycle 18 Day 1 | 7.0 (NA) — Number analyzed is 1 so SD is not available. | -3.3 (2.89) |
  Change at Cycle 19 Day 1: number analyzed (Participants) | 1 | 2 | 0
  Change at Cycle 19 Day 1 | 8.0 (NA) — Number analyzed is 1 so SD is not available. | -5.5 (13.44) |
  Change at Cycle 20 Day 1: number analyzed (Participants) | 1 | 1 | 0
  Change at Cycle 20 Day 1 | 8.0 (NA) — Number analyzed is 1 so SD is not available. | 2.0 (NA) — Number analyzed is 1 so SD is not available. |
  Change at Cycle 21 Day 1: number analyzed (Participants) | 1 | 1 | 0
  Change at Cycle 21 Day 1 | 8.0 (NA) — Number analyzed is 1 so SD is not available. | -5.0 (NA) — Number analyzed is 1 so SD is not available. |
  Change at Cycle 22 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Change at Cycle 22 Day 1 |  | -5.0 (NA) — Number analyzed is 1 so SD is not available. |
  Change at Cycle 23 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Change at Cycle 23 Day 1 |  | -5.0 (NA) — Number analyzed is 1 so SD is not available. |
  Change at End of Treatment: number analyzed (Participants) | 75 | 72 | 80
  Change at End of Treatment | -8.5 (17.40) | -8.0 (18.99) | -12.7 (21.34)
  Change at 30 Day Follow Up: number analyzed (Participants) | 24 | 16 | 21
  Change at 30 Day Follow Up | -11.1 (20.23) | -5.9 (20.18) | -11.0 (17.51)

44. Secondary Outcome: (Phase 3) Change From Baseline in the Participant Global Impression of Change (PGIC) in Triplet Arm vs Control Arm, Doublet Arm vs Control, and Triplet vs Doublet
Description: The PGIC is a measure of participant's perceptions of change in their symptoms over time that can be used as an anchoring method to determine the minimal clinically important difference for other participant reported outcome (PROs). For this assessment, participants answered the following question: "Since starting treatment, my colorectal cancer symptoms are: (1) very much improved, (2) much improved, (3) minimally improved, (4) no change, (5) minimally worse, (6) much worse or (7) very much worse."
Time Frame: as for outcome 42
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Phase 3: Triplet Arm | Phase 3:Doublet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 224 | 220 | 221
Units on a scale
  Baseline: number analyzed (Participants) | 153 | 152 | 149
  Baseline | 3.8 (1.30) | 3.8 (1.30) | 3.9 (1.28)
  Change at Cycle 1 Day 1: number analyzed (Participants) | 91 | 92 | 83
  Change at Cycle 1 Day 1 | -0.1 (0.93) | 0.1 (1.21) | 0.0 (0.90)
  Change at Cycle 2 Day 1: number analyzed (Participants) | 127 | 130 | 90
  Change at Cycle 2 Day 1 | -0.7 (1.44) | -0.8 (1.60) | -0.3 (1.52)
  Change at Cycle 3 Day 1: number analyzed (Participants) | 101 | 105 | 37
  Change at Cycle 3 Day 1 | -0.9 (1.44) | -1.2 (1.53) | -0.5 (1.56)
  Change at Cycle 4 Day 1: number analyzed (Participants) | 80 | 79 | 28
  Change at Cycle 4 Day 1 | -0.9 (1.49) | -1.1 (1.68) | -0.5 (1.35)
  Change at Cycle 5 Day 1: number analyzed (Participants) | 66 | 59 | 19
  Change at Cycle 5 Day 1 | -0.9 (1.61) | -1.1 (1.69) | -0.7 (1.41)
  Change at Cycle 6 Day 1: number analyzed (Participants) | 45 | 40 | 9
  Change at Cycle 6 Day 1 | -0.8 (1.31) | -1.2 (1.70) | -0.8 (1.39)
  Change at Cycle 7 Day 1: number analyzed (Participants) | 30 | 36 | 7
  Change at Cycle 7 Day 1 | -1.1 (1.44) | -1.0 (1.61) | -1.1 (1.07)
  Change at Cycle 8 Day 1: number analyzed (Participants) | 23 | 27 | 5
  Change at Cycle 8 Day 1 | -1.2 (1.56) | -1.1 (1.58) | -1.0 (0.71)
  Change at Cycle 9 Day 1: number analyzed (Participants) | 21 | 21 | 5
  Change at Cycle 9 Day 1 | -0.8 (1.26) | -0.9 (1.37) | -1.0 (0.71)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 15 | 17 | 3
  Change at Cycle 10 Day 1 | -0.5 (1.51) | -0.6 (1.28) | -0.3 (0.58)
  Change at Cycle 11 Day 1: number analyzed (Participants) | 13 | 13 | 2
  Change at Cycle 11 Day 1 | -0.9 (1.38) | -1.1 (1.38) | 0.0 (0.00)
  Change at Cycle 12 Day 1: number analyzed (Participants) | 11 | 12 | 2
  Change at Cycle 12 Day 1 | -0.9 (1.45) | -0.8 (1.36) | -0.5 (0.71)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 8 | 10 | 1
  Change at Cycle 13 Day 1 | -1.3 (1.39) | -0.9 (1.52) | -1.0 (NA) — Number analyzed is 1 so SD is not available.
  Change at Cycle 14 Day 1: number analyzed (Participants) | 7 | 6 | 0
  Change at Cycle 14 Day 1 | -1.1 (1.46) | -1.5 (1.05) |
  Change at Cycle 15 Day 1: number analyzed (Participants) | 6 | 5 | 0
  Change at Cycle 15 Day 1 | -1.2 (1.47) | -1.6 (0.89) |
  Change at Cycle 16 Day 1: number analyzed (Participants) | 4 | 3 | 0
  Change at Cycle 16 Day 1 | -2.0 (0.82) | -0.7 (1.53) |
  Change at Cycle 17 Day 1: number analyzed (Participants) | 3 | 3 | 0
  Change at Cycle 17 Day 1 | -1.3 (1.53) | -1.0 (1.00) |
  Change at Cycle 18 Day 1: number analyzed (Participants) | 1 | 3 | 0
  Change at Cycle 18 Day 1 | -2.0 (NA) — Number analyzed is 1 so SD is not available. | -1.0 (1.00) |
  Change at Cycle 19 Day 1: number analyzed (Participants) | 1 | 2 | 0
  Change at Cycle 19 Day 1 | -3.0 (NA) — Number analyzed is 1 so SD is not available. | -0.5 (2.12) |
  Change at Cycle 20 Day 1: number analyzed (Participants) | 1 | 1 | 0
  Change at Cycle 20 Day 1 | -3.0 (NA) — Number analyzed is 1 so SD is not available. | -2.0 (NA) — Number analyzed is 1 so SD is not available. |
  Change at Cycle 21 Day 1: number analyzed (Participants) | 1 | 1 | 0
  Change at Cycle 21 Day 1 | -3.0 (NA) — Number analyzed is 1 so SD is not available. | -2.0 (NA) — Number analyzed is 1 so SD is not available. |
  Change at Cycle 22 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Change at Cycle 22 Day 1 |  | -2.0 (NA) — Number analyzed is 1 so SD is not available. |
  Change at Cycle 23 Day 1: number analyzed (Participants) | 0 | 1 | 0
  Change at Cycle 23 Day 1 |  | -2.0 (NA) — Number analyzed is 1 so SD is not available. |
  Change at End of Treatment: number analyzed (Participants) | 52 | 54 | 63
  Change at End of Treatment | 0.3 (1.85) | 0.1 (1.82) | 0.4 (1.58)
  Change at 30 Day Follow Up: number analyzed (Participants) | 18 | 10 | 19
  Change at 30 Day Follow Up | -0.1 (2.08) | 0.5 (1.43) | 0.7 (1.34)

45. Secondary Outcome: (Safety Lead-in) Evaluation of the Area Under the Concentration-Time Curve From Zero to the Last Measurable Time Point (AUClast) for Cetuximab
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: The pharmacokinetics (PK) set included all participants in the Safety Set who had at least 1 post-dose blood collection for PK with associated bioanalytical results. Participants were analyzed according to the actual treatment and dose received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter *hour
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Nanogram/milliliter *hour
  Cycle 1: number analyzed (Participants) | 34
  Cycle 1 | 841000 (22.2)
  Cycle 2: number analyzed (Participants) | 32
  Cycle 2 | 970000 (20.6)

46. Secondary Outcome: (Safety Lead-in) Evaluation of the Area Under the Concentration-Time Curve From Zero to the Last Measurable Time Point (AUClast) for Encorafenib
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: The PK set included all participants in the Safety Set who had at least 1 post-dose blood collection for PK with associated bioanalytical results. Participants were analyzed according to the actual treatment and dose received. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter *hour
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Nanogram/milliliter *hour
  Cycle 1: number analyzed (Participants) | 34
  Cycle 1 | 11300 (61.5)
  Cycle 2: number analyzed (Participants) | 29
  Cycle 2 | 6660 (61.7)

47. Secondary Outcome: (Safety Lead-in) Evaluation of the Area Under the Concentration-Time Curve From Zero to the Last Measurable Time Point (AUClast) for Binimetinib
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: as for outcome 46
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter *hour
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Nanogram/milliliter *hour
  Cycle 1: number analyzed (Participants) | 34
  Cycle 1 | 1960 (43.6)
  Cycle 2: number analyzed (Participants) | 29
  Cycle 2 | 1540 (44.7)

48. Secondary Outcome: (Safety Lead-in) Evaluation of the Area Under the Concentration-time Curve From Zero to the Last Measurable Time Point (AUClast) for Metabolite of Binimetinib (AR00426032)
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: as for outcome 46
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter *hour
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Nanogram/milliliter *hour
  Cycle 1: number analyzed (Participants) | 35
  Cycle 1 | 206 (46.7)
  Cycle 2: number analyzed (Participants) | 26
  Cycle 2 | 70.0 (95.5)

49. Secondary Outcome: (Safety Lead-in) Evaluation of the Maximum Concentration (Cmax) for Cetuximab
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: as for outcome 46
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Nanogram/milliliter
  Cycle 1: number analyzed (Participants) | 34
  Cycle 1 | 195000 (22.2)
  Cycle 2: number analyzed (Participants) | 32
  Cycle 2 | 199000 (26.8)

50. Secondary Outcome: (Safety Lead-in) Evaluation of the Maximum Concentration (Cmax) for Encorafenib
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: as for outcome 46
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Nanogram/milliliter
  Cycle 1: number analyzed (Participants) | 34
  Cycle 1 | 3360 (65.1)
  Cycle 2: number analyzed (Participants) | 29
  Cycle 2 | 2490 (75.6)

51. Secondary Outcome: (Safety Lead-in) Evaluation of the Maximum Concentration (Cmax) for Binimetinib
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: as for outcome 46
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Nanogram/milliliter
  Cycle 1: number analyzed (Participants) | 35
  Cycle 1 | 654 (50.8)
  Cycle 2: number analyzed (Participants) | 26
  Cycle 2 | 524 (70.1)

52. Secondary Outcome: (Safety Lead-in) Evaluation of the Maximum Concentration (Cmax) for Metabolite of Binimetinib (AR00426032)
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: as for outcome 46
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Nanogram/milliliter
  Cycle 1: number analyzed (Participants) | 35
  Cycle 1 | 59.9 (50.8)
  Cycle 2: number analyzed (Participants) | 26
  Cycle 2 | 20.5 (119)

53. Secondary Outcome: (Safety Lead-in) Evaluation of the Time of Maximum Observed Concentration (Tmax) for Cetuximab
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: as for outcome 46
Measure: Median (Full Range); unit: Hours
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Hours
  Cycle 1: number analyzed (Participants) | 34
  Cycle 1 | 3.77 [1.83 to 6.05]
  Cycle 2: number analyzed (Participants) | 32
  Cycle 2 | 3.05 [1.00 to 6.17]

54. Secondary Outcome: (Safety Lead-in) Evaluation of the Time of Maximum Observed Concentration (Tmax) for Encorafenib
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: as for outcome 46
Measure: Median (Full Range); unit: Hours
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Hours
  Cycle 1: number analyzed (Participants) | 34
  Cycle 1 | 2.00 [.883 to 6.25]
  Cycle 2: number analyzed (Participants) | 29
  Cycle 2 | 2.00 [.950 to 5.73]

55. Secondary Outcome: (Safety Lead-in) Evaluation of the Time of Maximum Observed Concentration (Tmax) for Binimetinib
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: as for outcome 46
Measure: Median (Full Range); unit: Hours
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Hours
  Cycle 1: number analyzed (Participants) | 35
  Cycle 1 | 1.98 [.883 to 5.67]
  Cycle 2: number analyzed (Participants) | 26
  Cycle 2 | 1.04 [.900 to 4.00]

56. Secondary Outcome: (Safety Lead-in) Evaluation of the Time of Maximum Observed Concentration (Tmax) for Metabolite of Binimetinib (AR00426032)
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: as for outcome 46
Measure: Median (Full Range); unit: Hours
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Hours
  Cycle 1: number analyzed (Participants) | 35
  Cycle 1 | 2.00 [.833 to 5.78]
  Cycle 2: number analyzed (Participants) | 26
  Cycle 2 | 1.58 [.933 to 6.52]

57. Secondary Outcome: (Safety Lead-in) Evaluation of the Steady-State Concentration Measured Just Before the Next Dose of Study Drug (Ctrough) for Binimetinib
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: The PK set included all participants in the Safety Set who had at least 1 post-dose blood collection for PK with associated bioanalytical results. Participants were analyzed according to the actual treatment and dose received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Nanogram/milliliter | 55.3 (61.5)

58. Secondary Outcome: (Safety Lead-in) Evaluation of the Steady-State Concentration Measured Just Before the Next Dose of Study Drug (Ctrough) for Encorafenib
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: as for outcome 57
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Nanogram/milliliter | 18.9 (191)

59. Secondary Outcome: (Safety Lead-in) Evaluation of the Steady-State Concentration Measured Just Before the Next Dose of Study Drug (Ctrough) for Cetuximab
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: as for outcome 57
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Nanogram/milliliter | 55400 (54.8)

60. Secondary Outcome: (Safety Lead-in) Evaluation of the Steady-State Concentration Measured Just Before the Next Dose of Study Drug (Ctrough) for a Metabolite of Binimetinib
Time Frame: Predose and 1, 2, 4 and 6 hours post-dose on Day 1 of Cycles 1 and 2 (each cycle of 28 days)
Population: as for outcome 57
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Combined Safety Lead-in
Number analyzed (Participants) | 37
Nanogram/milliliter | 3.41 (68.5)

61. Secondary Outcome: (Phase 3) Evaluation of the Model-Based Oral Clearance (CL/F) for Encorafenib
Description: The reported cross-arm CL/F value is a fixed-effect parameter determined from a population PK analysis. The analysis included pooled data from participants enrolled in multiple studies including those who were not enrolled in this study. The NCTID include: NCT01719380, NCT01543698, and NCT01436656. An additional study ARRAY-162-105 is not required to register.
Time Frame: 2 and 6 hours post-dose on Day 1 of Cycle 1, Predose and 2 hours post-dose on Day 1 of Cycle 2 (each cycle of 28 days)
Population: The analysis set included all participants in the PK set with measurable plasma concentrations of the test drug plus concentrations from subjects from 4 additional clinical studies. Participants were analyzed according to the actual treatment and dose received.
Measure: Geometric Mean (95% Confidence Interval); unit: Liter/hour
Groups:
- Pharmacokinetic Population of Encorafenib: Encorafenib + binimetinib + cetuximab. Encorafenib + cetuximab. Investigator's choice of either irinotecan/cetuximab or FOLFIRI/cetuximab.
Arm/Group | Pharmacokinetic Population of Encorafenib
Number analyzed (Participants) | 394
Liter/hour | 16.4 [14.9 to 17.5]

62. Secondary Outcome: (Phase 3) Evaluation of the Model-Based Oral Clearance (CL/F) for Binimetinib
Description: as for outcome 61
Time Frame: 2 and 6 hours post-dose on Day 1 of Cycle 1, Predose and 2 hours post-dose on Day 1 of Cycle 2 (each cycle of 28 days)
Population: as for outcome 61
Measure: Geometric Mean (95% Confidence Interval); unit: Liter/hour
Arm/Group | Pharmacokinetic Population of Encorafenib
Number analyzed (Participants) | 181
Liter/hour | 19.0 [17.7 to 20.6]

63. Secondary Outcome: (Phase 3) Evaluation of the Model-Based Clearance (CL) for Cetuximab
Description: as for outcome 61
Time Frame: 2 and 6 hours post-dose on Day 1 of Cycle 1, Predose and 2 hours post-dose on Day 1 of Cycle 2 (each cycle of 28 days)
Population: as for outcome 61
Measure: Geometric Mean (95% Confidence Interval); unit: Liter/hour
Arm/Group | Pharmacokinetic Population of Encorafenib
Number analyzed (Participants) | 261
Liter/hour | 0.0154 [0.0114 to 0.0225]

64. Secondary Outcome: Phase 3: Number of Participants With Clinically Notable Shifts in Hematology and Coagulation Laboratory Parameters
Description: Clinically notable shifts was defined as worsening by at least 2 grades or to more than or equal to (>=) Grade 3 based on Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 where Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life threatening and Grade 5: death.
Time Frame: From start of study treatment until 30 days post last dose of study treatment (for triplet arm: maximum treatment exposure of 277.4 weeks; for doublet arm: maximum treatment exposure of 268 weeks; for Control arm: maximum treatment exposure of 108 weeks)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Triplet Arm | Phase 3: Doublet Arm | Phase 3:Control Arm
Number analyzed (Participants) | 222 | 216 | 193
Participants
  Activated Partial Thromboplastin Time - Hyper | 9 | 9 | 4
  Hemoglobin - Hyper | 0 | 0 | 0
  Hemoglobin - Hypo | 97 | 30 | 17
  Leukocytes - Hyper | 0 | 0 | 0
  Leukocytes - Hypo | 2 | 9 | 51
  Lymphocytes - Hyper | 12 | 3 | 4
  Lymphocytes - Hypo | 25 | 47 | 57
  Neutrophils - Hypo | 4 | 8 | 65
  Platelets - Hypo | 1 | 5 | 4
  Prothrombin Intl. Normalized Ratio - Hyper | 3 | 2 | 2

65. Secondary Outcome: Phase 3: Number of Participants With Clinically Notable Shifts in Serum Chemistry Laboratory Parameters
Description: Clinically notable shifts was defined as worsening by at least 2 grades or to >= Grade 3 based on CTCAE version 4.03 where Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life threatening and Grade 5: death.
Time Frame: as for outcome 64
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Triplet Arm | Phase 3: Doublet Arm | Phase 3: Control Arm
Number analyzed (Participants) | 222 | 216 | 193
Participants
  Alanine Aminotransferase - Hyper | 11 | 7 | 10
  Albumin - Hypo | 50 | 16 | 17
  Alkaline Phosphatase - Hyper | 13 | 12 | 18
  Aspartate Aminotransferase - Hyper | 11 | 7 | 9
  Bilirubin - Hyper | 11 | 13 | 12
  Calcium - Hyper | 1 | 0 | 0
  Calcium - Hypo | 15 | 8 | 7
  Creatine Kinase - Hyper | 18 | 1 | 3
  Creatinine - Hyper | 45 | 11 | 6
  Glucose - Hyper | 8 | 16 | 4
  Glucose - Hypo | 4 | 0 | 1
  Magnesium - Hyper | 0 | 1 | 2
  Magnesium - Hypo | 11 | 4 | 9
  Potassium - Hyper | 14 | 10 | 5
  Potassium - Hypo | 5 | 7 | 9
  Sodium - Hyper | 1 | 1 | 2
  Sodium - Hypo | 10 | 4 | 5
  Troponin I - Hyper | 0 | 0 | 0
  Urate - Hyper | 4 | 2 | 1

66. Secondary Outcome: Phase 3: Number of Participants With Clinically Notable Shifts in Urinalysis Laboratory Parameters
Description: as for outcome 65
Time Frame: as for outcome 64
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Triplet Arm | Phase 3: Doublet Arm | Phase 3: Control Arm
Number analyzed (Participants) | 222 | 216 | 193
Participants | 8 | 8 | 5

67. Secondary Outcome: Phase 3: Number of Participants With Newly Occurring Clinically Notable Vital Sign Abnormalities
Description: Newly occurring clinically notable changes was defined as participants not meeting the criterion at baseline and meeting criterion post-baseline. The criterion included: low/high systolic blood pressure (SBP): <= 90 millimeters of mercury (mmHg) with decrease from baseline of >= 20mmHg or >= 160mmHg with increase from baseline of >= 20mmHg, low or high diastolic blood pressure (DBP): <= 50mmHg with decrease from baseline of >= 15mmHg or >= 100mmHg with increase from baseline of >= 15mmHg, low or high pulse: <= 50 beats/min with decrease from baseline of >= 15 beats/min or >= 120 beats/min with increase from baseline of >= 15 beats/min, low or high temperature: <= 36 degree Celsius (deg C) or >= 37.5 deg C.
Time Frame: as for outcome 64
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Triplet Arm | Phase 3: Doublet Arm | Phase 3: Control Arm
Number analyzed (Participants) | 222 | 216 | 193
Participants
  Diastolic Blood Pressure - High | 8 | 6 | 7
  Diastolic Blood Pressure - Low | 21 | 27 | 5
  Pulse Rate - High | 23 | 14 | 20
  Pulse Rate - Low | 3 | 4 | 3
  Systolic Blood Pressure - High | 19 | 13 | 5
  Systolic Blood Pressure - Low | 37 | 28 | 10
  Temperature - High | 33 | 23 | 25
  Temperature - Low | 93 | 84 | 55

68. Secondary Outcome: Phase 3: Number of Participants With Newly Occurring Clinically Notable Electrocardiogram (ECG) Values
Description: Newly occurring clinically notable changes was defined as participants not meeting the criterion at baseline and meeting criterion post-baseline. The criterion included: heart rate- decrease from baseline > 25% and to a value < 50 and increase from baseline > 25% and to a value > 100. QT interval- new > 450 (millisecond) msec, new > 480 msec, new > 500 msec, increase from baseline > 30 msec and increase from baseline > 60 msec. QTcF- new > 450 msec, new > 480 msec, new > 500 msec, increase from baseline > 30 msec and increase from baseline > 60 msec.
Time Frame: as for outcome 64
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Triplet Arm | Phase 3: Doublet Arm | Phase 3: Control Arm
Number analyzed (Participants) | 222 | 216 | 193
Participants
  Heart Rate - Decrease from baseline > 25% and to a value < 50 | 1 | 4 | 0
  Heart Rate - Increase from baseline > 25% and to a value > 100 | 27 | 24 | 28
  QT Interval - New > 450 millisecond (msec) | 17 | 30 | 7
  QT Interval - New > 480 msec | 4 | 7 | 2
  QT Interval - New > 500 msec | 3 | 5 | 0
  QT Interval - increase from baseline > 30 msec | 97 | 99 | 32
  QT Interval - increase from baseline > 60 msec | 22 | 21 | 10
  QTcF - New > 450 msec | 39 | 51 | 23
  QTcF - New > 480 msec | 9 | 18 | 5
  QTcF - New > 500 msec | 1 | 6 | 2
  QTcF - increase from baseline > 30 msec | 59 | 75 | 24
  QTcF - increase from baseline > 60 msec | 12 | 20 | 5

69. Secondary Outcome: Phase 3: Number of Participants With Shift in Visual Acuity Logarithm of the Minimum Angle of Resolution (LogMAR) Score
Description: Visual acuity was measured using the Snellen visual acuity conversion chart. This was determined by establishing the smallest optotypes that could be identified correctly by the participant at a given observation distance. Snellen visual acuity was reported as a Snellen fraction (m/M) in which the numerator (m) indicated the test distance and the denominator (M) indicated the distance at which the gap of the equivalent Landolt ring subtends 1 minute of arc. The LogMAR score was calculated as - log(m/M). The maximum increase in score of <= 0, 0 to < 0.1, 0.1 to < 0.2, 0.2 to < 0.3 and >=0.3 relative to baseline in LogMAR were reported in this endpoint.
Time Frame: as for outcome 64
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Triplet Arm | Phase 3: Doublet Arm | Phase 3: Control Arm
Number analyzed (Participants) | 222 | 216 | 193
Participants
  Baseline <=0 to >0-<0.1 | 33 | 8 | 0
  Baseline <=0 to 0.1-<0.2 | 15 | 3 | 0
  Baseline <=0 to 0.2-<0.3 | 4 | 0 | 0
  Baseline <=0 to >=0.3 | 6 | 1 | 0
  Baseline <=0 to missing score | 9 | 86 | 129
  Baseline >0-<0.1 to <=0 | 17 | 6 | 0
  Baseline >0-<0.1 to 0.1-<0.2 | 7 | 2 | 0
  Baseline >0-<0.1 to 0.2-<0.3 | 4 | 1 | 0
  Baseline >0-<0.1 to >=0.3 | 3 | 0 | 0
  Baseline >0-<0.1 to missing score | 3 | 25 | 30
  Baseline 0.1-<0.2 to <=0 | 5 | 1 | 0
  Baseline 0.1-<0.2 to >0-<0.1 | 1 | 0 | 0
  Baseline 0.2-<0.3 to <=0 | 1 | 0 | 0
  Baseline 0.2-<0.3 to >0-<0.1 | 3 | 0 | 0
  Baseline 0.2-<0.3 to 0.1-<0.2 | 3 | 1 | 0
  Baseline 0.2-<0.3 to missing score | 1 | 4 | 5
  Baseline >=0.3 to <=0 | 9 | 2 | 0
  Baseline >=0.3 to >0-<0.1 | 4 | 0 | 0
  Baseline >=0.3 to 0.1-<0.2 | 1 | 1 | 0
  Baseline >=0.3 to 0.2-<0.3 | 2 | 0 | 0
  Baseline >=0.3 to missing score | 1 | 19 | 13
  Baseline 0.1-<0.2 to 0.2-<0.3 | 0 | 3 | 0
  Baseline 0.1-<0.2 to missing score | 0 | 9 | 7

70. Secondary Outcome: Phase 3: Number of Participants With Shifts in Left Ventricular Ejection Fraction (LVEF) From Baseline to Maximum Grade On-treatment
Description: Left ventricular ejection fraction (LVEF) abnormalities were defined according to CTCAE version 4.03 where Grade 0: Non-missing value below Grade 2, Grade 2: LVEF between 40% and 50% or absolute change from baseline between -10% and < -20%, Grade 3: LVEF between 20% and 39% or absolute change from baseline <= -20%, Grade 4: LVEF lower than 20%. Categories with at least 1 non-zero data values showing any shift in Grade from baseline to 1 day after dose 1 (post-baseline) were reported. Participants whose grade category was unchanged (e.g. Grade 0 to Grade 0) were not reported.
Time Frame: as for outcome 64
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 3: Triplet Arm | Phase 3: Doublet Arm | Phase 3: Control Arm
Number analyzed (Participants) | 222 | 216 | 193
Participants
  Baseline Grade 0 to Grade 2 post baseline | 27 | 0 | 0
  Baseline Grade 0 to Grade 3 post baseline | 1 | 1 | 0
  Baseline Grade 0 to missing grade | 17 | 205 | 186
  Baseline Grade 2 to missing grade | 0 | 3 | 2
  Baseline missing grade to Grade 0 post baseline | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) were collected from initiation of study drug through 30 days after the last dose of study drug. For CSLI: maximum treatment exposure of 280 weeks; for Phase 3- Triplet arm: maximum treatment exposure of 277.4 weeks; for Phase 3- Doublet arm: maximum treatment exposure of 268 weeks; for Phase 3- Control arm: maximum treatment exposure of 108 weeks
Description: An AE is defined as the appearance of (or worsening of any pre-existing) undesirable signs, symptoms, or medical conditions that occur after participant's signed informed consent has been obtained. For non-SAEs and SAEs: safety set consisted of all participants who received at least 1 dose of study drug and had at least 1 post-treatment assessment, which may have included death. For all-cause mortality: FAS for the Phase 3 portion of the study consisted of all randomized Phase 3 participants.
Arm/Group | Combined Safety Lead-in | Phase 3: Triplet Arm | Phase 3: Doublet Arm | Phase 3: Control Arm
All-Cause Mortality (participants affected / at risk) | 30/37 | 209/224 | 193/220 | 198/221
Serious Adverse Events (participants affected / at risk) | 22/37 | 118/222 | 91/216 | 78/193
Other Adverse Events (participants affected / at risk) | 36/37 | 218/222 | 212/216 | 187/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Safety Lead-in (N=37) | Phase 3: Triplet Arm (N=222) | Phase 3: Doublet Arm (N=216) | Phase 3: Control Arm (N=193)
Diarrhoea (Gastrointestinal disorders) | 1 | 10 | 0 | 10
Vomiting (Gastrointestinal disorders) | 2 | 6 | 2 | 4
Anaemia (Blood and lymphatic system disorders) | 1 | 6 | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 5 | 4 | 4
Intestinal obstruction (Gastrointestinal disorders) | 0 | 11 | 12 | 7
Large intestine perforation (Gastrointestinal disorders) | 1 | 3 | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 2 | 4
Hepatic failure (Hepatobiliary disorders) | 0 | 3 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 5 | 3 | 3
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3
Pulmonary embolism (Blood and lymphatic system disorders) | 1 | 8 | 3 | 5
Acute kidney injury (Renal and urinary disorders) | 1 | 8 | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 7 | 5 | 4
Bacteraemia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 1
Bile duct obstruction (Gastrointestinal disorders) | 0 | 2 | 3 | 2
Urinary tract infection (Renal and urinary disorders) | 4 | 2 | 5 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 5 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 4 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 5
Infusion-related reaction (Blood and lymphatic system disorders) | 5 | 1 | 7 | 6
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 6 | 4 | 4
Colitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Abdominal distention (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
intestinal perforation (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestine ulcer (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 1 | 1 | 0
Cholangitis infective (Infections and infestations) | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 1 | 0
Gastrintestinal infection (Infections and infestations) | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 2 | 0
Wound abscess (Infections and infestations) | 0 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 1 | 1 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 2 | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 2 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 1 | 1
Death (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 1 | 3
Asthenia (General disorders) | 0 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestinal ulcer hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 7 | 3 | 1
Oesophageal ulcer hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 4 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Tumor haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 2 | 3 | 2
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 1
Abdominal infection (Infections and infestations) | 0 | 2 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 4 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 4 | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 2 | 0 | 0 | 0
Infectious colitis (Infections and infestations) | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 3 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 3 | 1 | 2
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 2 | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Streptococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 5 | 6 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 8 | 3 | 5
Prerenal failure (Renal and urinary disorders) | 0 | 2 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 4 | 1 | 0
Catheter site thrombosis (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 2 | 0
General physical health deterioration (General disorders) | 0 | 1 | 1 | 2
Malaise (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Perforation (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 5 | 2 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0
Device occlusion (Product Issues) | 1 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1 | 3 | 2
Radiation inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Periostitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 2 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Analgesic therapy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Esophageal ulcer hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Safety Lead-in (N=37) | Phase 3: Triplet Arm (N=222) | Phase 3: Doublet Arm (N=216) | Phase 3: Control Arm (N=193)
Diarrhoea (Gastrointestinal disorders) | 29 | 150 | 85 | 96
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 25 | 113 | 65 | 77
Nausea (Gastrointestinal disorders) | 22 | 107 | 80 | 84
Vomiting (Gastrointestinal disorders) | 19 | 99 | 58 | 59
Anaemia (Blood and lymphatic system disorders) | 16 | 105 | 44 | 37
Fatigue (General disorders) | 20 | 74 | 74 | 54
Abdominal pain (Gastrointestinal disorders) | 14 | 74 | 60 | 54
Decreased appetite (Metabolism and nutrition disorders) | 15 | 67 | 68 | 56
Asthenia (General disorders) | 6 | 63 | 51 | 52
Constipation (Gastrointestinal disorders) | 14 | 64 | 39 | 39
Dry Skin (Skin and subcutaneous tissue disorders) | 19 | 49 | 28 | 17
Pyrexia (General disorders) | 16 | 53 | 43 | 30
Rash (Skin and subcutaneous tissue disorders) | 3 | 49 | 35 | 28
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 35 | 24 | 10
Back Pain (Musculoskeletal and connective tissue disorders) | 8 | 36 | 32 | 27
Vision blurred (Eye disorders) | 12 | 27 | 10 | 1
Weight decreased (Investigations) | 3 | 25 | 26 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 26 | 52 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 26 | 22 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 29 | 28 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 23 | 35 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 22 | 30 | 20
Headache (Nervous system disorders) | 7 | 21 | 43 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 16 | 14 | 25
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 19 | 26 | 2
Insomnia (Psychiatric disorders) | 2 | 15 | 25 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 12 | 32 | 5
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 4 | 36
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 34 | 0
Neutrophil count decreased (Investigations) | 0 | 2 | 1 | 21
Abdominal pain upper (Gastrointestinal disorders) | 5 | 24 | 22 | 15
Dyspepsia (Gastrointestinal disorders) | 4 | 18 | 9 | 7
Flatulence (Gastrointestinal disorders) | 0 | 15 | 6 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 21 | 6 | 1
Dry Mouth (Gastrointestinal disorders) | 2 | 11 | 10 | 8
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 10 | 6 | 6
Abdominal distension (Gastrointestinal disorders) | 2 | 10 | 16 | 8
Intestinal obstruction (Gastrointestinal disorders) | 0 | 11 | 12 | 7
Palmar-planar erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 6 | 31 | 11 | 15
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 19 | 19 | 11
Skin fissures (Skin and subcutaneous tissue disorders) | 9 | 21 | 9 | 13
Erythema (Skin and subcutaneous tissue disorders) | 2 | 9 | 13 | 4
Eczema (Skin and subcutaneous tissue disorders) | 2 | 5 | 2 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 1 | 16 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 17 | 3
Chills (General disorders) | 6 | 15 | 6 | 3
Malaise (General disorders) | 7 | 5 | 6 | 11
Urinary tract infection (Infections and infestations) | 7 | 26 | 16 | 5
Paronychia (Infections and infestations) | 6 | 21 | 13 | 20
Rash pustular (Infections and infestations) | 6 | 13 | 4 | 4
Conjunctivitis (Infections and infestations) | 2 | 16 | 12 | 3
Cystitis (Infections and infestations) | 2 | 6 | 2 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 20 | 6 | 6
Dizziness (Nervous system disorders) | 8 | 16 | 16 | 16
Neuropathy peripheral (Nervous system disorders) | 1 | 13 | 11 | 5
Dysgeusia (Nervous system disorders) | 6 | 11 | 10 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 7 | 5 | 4
Blood creatine phosphokinase increased (Investigations) | 11 | 26 | 3 | 4
Blood creatine increased (Investigations) | 11 | 25 | 6 | 1
Alanine aminotransferase increased (Investigations) | 6 | 16 | 15 | 14
Aspartate aminotransferase increased (Investigations) | 7 | 14 | 7 | 14
Ejection fraction decreased (Investigations) | 5 | 8 | 0 | 0
Blood bilirubin increased (Investigations) | 3 | 5 | 9 | 8
White blood cell count decrease (Investigations) | 0 | 2 | 2 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 22 | 5 | 4
Dry eye (Eye disorders) | 5 | 9 | 11 | 3
Retinal detachment (Eye disorders) | 2 | 6 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 8 | 16 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 12 | 3
Rhinnorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 6 | 1
Haematuria (Renal and urinary disorders) | 2 | 16 | 6 | 4
Hypotension (Vascular disorders) | 3 | 9 | 9 | 3
Hypertension (Vascular disorders) | 4 | 8 | 8 | 6
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 5 | 18 | 13
Depression (Psychiatric disorders) | 2 | 5 | 5 | 1
Palpitations (Cardiac disorders) | 2 | 3 | 4 | 1
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 1 | 1
Anal haemorrhage (Gastrointestinal disorders) | 2 | 6 | 1 | 2
Ascites (Gastrointestinal disorders) | 2 | 5 | 2 | 4
Colitis (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 6 | 32 | 13 | 45
Abdominal pain lower (Gastrointestinal disorders) | 2 | 5 | 4 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 6 | 10 | 21
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 12 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 3 | 4 | 5 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 4 | 3 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 6 | 12 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 10 | 5 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 7 | 3 | 4
Iron deficiency (Metabolism and nutrition disorders) | 3 | 2 | 3 | 1
Nasopharyngitis (Infections and infestations) | 3 | 12 | 15 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 9 | 10
Oedema peripheral (General disorders) | 6 | 30 | 24 | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 7 | 5 | 2
Chorioretinopathy (Eye disorders) | 2 | 3 | 0 | 0
Macular oedema (Eye disorders) | 3 | 1 | 1 | 0
Trichiasis (Eye disorders) | 4 | 1 | 0 | 0
Trichomegaly (Eye disorders) | 2 | 6 | 1 | 0
Visual impairment (Eye disorders) | 3 | 4 | 5 | 0
Vitreous floaters (Eye disorders) | 4 | 3 | 4 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 6 | 7 | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 1
Nervous system disorder (Nervous system disorders) | 2 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 2 | 1 | 10 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 15 | 0
Pollakiuria (Renal and urinary disorders) | 4 | 4 | 8 | 0
Proteinuria (Renal and urinary disorders) | 3 | 5 | 6 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 1 | 5 | 2
Wound (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT02928224/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT02928224/SAP_002.pdf